## **Statistical Analysis Plan**

A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy/Potency of a Single Dose of Xisomab 3G3, Administered at the Beginning of a Regular Hemodialysis Procedure, in Patients with End-Stage R14.3.5.3enal Disease on Chronic Hemodialysis

Protocol No: 3G3-18-02 Final Protocol Date: 25 May 2018 Amendment One Date: 14 June 2018

Compound Name: xisomab 3G3

Celerion Project CA23900 Final Version 1.0 Date: 20 December 2018

Aronora, Inc. 4640 SW Macadam Avenue, Ste 200A Portland, Oregon 97239, USA

Celerion 621 Rose Street, Lincoln, Nebraska 68502, USA 100 Alexis-Nihon Boulevard, Suite 360, Montreal, QC, H4M 2N8, Canada

## Statistical Analysis Plan Signature Page

| Compound | Name: xisomab 3G3 | |
|---|---|---|
| Protocol: 3 | G3-18-02 | |
| Study Title | e: A Phase 2, Randomized, Double-Blind, Place<br>and Efficacy/Potency of a Single Dose of Xise<br>Beginning of a Regular Hemodialysis Procedu<br>Renal Disease on Chronic Hemodialysis | omab 3G3, Administered at the |
| Issue Date: | 20 December 2018 | |
| Signature:_ | Mohammad Abu-Rashid, BPharm, MPhil<br>Senior Scientist, Clinical Pharmacology & Pha<br>Data Management and Biometrics, Celerion<br>100 Alexis Nihon Blvd., Suite 360<br>Montreal, Quebec H4M 2N8, Canada | Date: |
| ] | Nancy Wang, PhD Associate Director, Biostatistics Data Management and Biometrics, Celerion Lincoln, Nebraska, USA | Date: |
| Signature:_ | Christina Lorentz, PhD Senior Scientist Aronora, Inc. Portland, Oregon 97239, USA | Date: |

## **Table of Contents**

| 1. | INT | RODUCTION | 5 |
|---|---|---|---|
| 2. | OBJ | ECTIVES AND ENDPOINTS | 5 |
| | 2.1 | Objectives | |
| | 2.2 | Endpoints | |
| 3. | STU | JDY DESIGN | 6 |
| <i>4</i> . | | ALYSIS POPULATIONS | |
| т. | 4.1 | Analysis Populations | |
| | 4.2 | Preliminary Data and Interim Analysis | |
| 5. | | EATMENT DESCRIPTIONS | |
| 6. | | ARMACOKINETIC ANALYSIS | |
| 0. | 6.1 | Measurements and Collection Schedule | |
| | 6.2 | Bioanalytical Method | |
| | 6.3 | Investigational Product and PK Analyte Information | |
| | | 6.3.1 Xisomab 3G3 | |
| | 6.4 | Pharmacokinetic Concentrations | |
| | 6.5 | Noncompartmental Pharmacokinetic Analysis and Parameter Calculation | 9 |
| | | 6.5.1 Plasma Pharmacokinetic Parameters | 9 |
| | 6.6 | Data Summarization and Presentation of PK Parameters | 11 |
| 7. | PHA | ARMACODYNAMICS | 12 |
| | 7.1 | Pharmacodynamic Assessment | 12 |
| | | 7.1.1 Drug potency | 12 |
| | | 7.1.2 Efficiency of HD | 12 |
| | 7.2 | Data Summarization and Presentation of PD Parameters | 13 |
| | | 7.2.1 aPTT 13 | |
| | | 7.2.2 BUN and Potassium: | 14 |
| | | 7.2.3 URR and KT/V | 14 |
| | | 7.2.4 Clotting in the Drip Chamber and Dialysis Filter | 15 |
| | | 7.2.5 Dialysate Analysis | |
| 8. | SAF | ETY | 15 |
| | 8.1 | Subject Discontinuation | |
| | 8.2 | Demographics | 16 |
| | 8.3 | Adverse Events | 16 |
| | 8.4 | Clinical Laboratory Tests (Serum Chemistry, Hematology, Coagulation | 14 |
| | 8.5 | and Urinalysis) | |
| | 8.6 | Electrocardiogram. | |
| | ~.~ | | / |

| | 0.7 | Concernitant Medications | 17 |
|-----|------|------------------------------------------------|----|
| | 8.7 | Concomitant Medications | |
| | 8.8 | Physical Examination | |
| | 8.9 | Vascular Access Site Reaction | 18 |
| | 8.10 | Bleeding Time | 18 |
| | | Medical History | |
| | | Immunogenecity | |
| 9. | SUM | MARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS | 18 |
| 10. | SUM | MARY TABLES AND FIGURES | 18 |
| | 10.1 | In-text Summary Tables and Figures | 19 |
| | | Section 14 Summary Tables and Figures | |
| | | Section 16 Data Listings | |
| 11. | TAB | LE AND FIGURE SHELLS | 29 |
| | 11.1 | In-text Summary Tables Shells | 30 |
| | | Figures Shells | |
| | | Section 14 Summary Tables Shells | |
| 12. | LIST | ING SHELLS | 69 |

#### 1. INTRODUCTION

The following statistical analysis plan (SAP) provides the framework for the summarization of the data from this study. The SAP may change due to unforeseen circumstances. Any changes made from the planned analysis within the protocol, after the unblinding, or locking of the database will be documented in the clinical study report (CSR). The section referred to as Table Shells within this SAP describes the traceability of the tables, figures, and listings (TFLs) back to the data. Note that the header for this page will be the one used for the main body of the CSR.

Any additional exploratory analyses not addressed within this statistical analysis plan (SAP) and/or driven by the data, or requested by Aronora Inc., will be considered out of scope and must be described in the CSR.

#### 2. OBJECTIVES AND ENDPOINTS

## 2.1 Objectives

The primary objective of the study is to assess the safety and tolerability of a single dose of xisomab 3G3 when injected through a port into the proximal (arterial) dialysis line immediately after initiation of a hemodialysis (HD) procedure in patients with end stage renal disease (ESRD).

The secondary objectives of the study are as follows:

- To assess the pharmacodynamics (PD) of a single dose of xisomab 3G3 when injected through a port into the proximal (arterial) dialysis line immediately after initiation of a HD procedure in patients with ESRD.
- To assess the efficacy of a single dose of xisomab 3G3 on HD efficiency when injected through a port into the proximal (arterial) dialysis line immediately after initiation of a HD procedure in patients with ESRD.
- To assess the pharmacokinetics (PK) of a single dose of xisomab 3G3 when injected through a port into the proximal (arterial) dialysis line immediately after initiation of a HD procedure in patients with ESRD.

## 2.2 Endpoints

#### **Primary outcome measures:**

• The safety and tolerability of xisomab 3G3 will be evaluated versus pre-treatment and placebo by reviewing number and severity of adverse events and use of concomitant medications, physical examination, vascular access site reaction, bleeding time, and changes in vital signs, ECGs, and clinical laboratory evaluations.

#### **Secondary outcome measures:**

- PD using dose-dependency of drug potency, determined by measuring changes in the coagulation parameter (aPTT), and thrombus accumulation (assessed and ranked by visual inspection) within the dialyzer cartridges and total protein accumulation in the HD filter after xisomab 3G3-treatment versus pre-treatment and placebo.
- Hemodialysis efficiency using blood urea nitrogen (BUN) and potassium levels will be measured before and after hemodialysis to calculate URR and Kt/V.

Note: Kt/V = volume of fluid completely cleared of urea [K = dialyzer clearance (mL/min), t = time of dialysis] and V = volume of water a patients body contains. Formulas to calculate Kt/V and URR are located under Section 7.2.3.

#### Other outcome measures:

- The following PK parameters will be calculated for xisomab 3G3 in plasma, as appropriate: AUC0-t, AUC0-inf, AUC%extrap, Cmax, Tmax, Kel, t½, CL, and Vss.
- Development of immunity or antibodies against xisomab 3G3 after drug exposure.

#### 3. STUDY DESIGN

This is a phase 2, randomized, double-blind, placebo-controlled, single-dose study of xisomab 3G3 designed to evaluate the safety, efficacy/potency, and PK at 2 dose levels administered to patients with ESRD undergoing HD.

Patients will be enrolled into Cohort 1 or Cohort 2; cohorts will be dosed sequentially. Within a cohort, patients will be randomized to active drug or placebo as summarized below:

| Cohort | Treatment | Active:Placebo | <b>Cohort Size</b> |
|---|---|---|---|
| 1 | Infusion dose of 0.25 mg/kg xisomab 3G3 or placebo | 2:1 | 9-12 |
| 2 | Infusion dose of 0.5 mg/kg xisomab 3G3 or placebo | 2:1 | 9-12 |

This study includes a screening period of 28 days prior to checking-in to the clinical research unit on Day -8. From Day -7 (one week prior to dosing on Day 1) through Day -1, all patients will undergo HD 3 times and will be assessed for all scheduled procedures and endpoints before and after each HD session.

On Study Day 1, prior to dosing, patients will undergo baseline measurements followed by initiation of a regular HD procedure, consistently using only one type of dialyzer cartridge in each patient. Immediately after the start of blood perfusion, a single dose of xisomab 3G3 or matching placebo will be injected through a port into the flowing arterial blood in the proximal dialysis line. Patients will continue to undergo HD procedures and scheduled assessments from Day 1 through Day 12.

Study assessments will include physical examinations, vital signs, electrocardiogram (ECGs), clinical laboratory tests, HD vascular access site (AV fistula or AV graft) reaction, antibody titer (immunogenicity), adverse events (AEs), PD blood sampling (coagulation parameters), and PK blood sampling to be performed throughout the study. On Days -7, -5, and -3 and Days 1, 3, 5, and 12, bleeding time from the HD vascular access sites on the AV fistula or AV graft (ladder or buttonhole technique) will be evaluated at the end of the HD session. The dialyzer cartridge will be rinsed and visually inspected at the end of the HD procedure and graded against a standardized visual assessment scale. After visual assessment, the used and rinsed dialyzer cartridge will be frozen and saved for later retained content (deposited blood-derived material) analysis. The number of dialyzer cartridges used for the HD session will be recorded.

All patients who received the study drug or placebo (including patients who terminate the study early) will undergo follow-up procedures at the Clinical Research Unit (CRU) approximately 12 days after dosing.

#### 4. ANALYSIS POPULATIONS

### 4.1 Analysis Populations

## **Safety Population**

The safety population will include all patients who received at least one dose of study drug (active or placebo).

### **Pharmacokinetic Population**

Samples from all patients receiving the active drug will be assayed even if the patients do not complete the study. All patients receiving the active drug who comply sufficiently with the protocol and display an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations) will be included in the statistical analyses.

#### Pharmacodynamic Population

All patients who received the study drug (active or placebo) and had at least one postdose measurement of any of the PD assessment will be included in the statistical analyses.

### 4.2 Preliminary Data and Interim Analysis

Celerion has not been contracted to complete any interim safety, PK, and PD analyses.

#### 5. TREATMENT DESCRIPTIONS

Patients will receive a single infusion dose of 0.25 mg/kg xisomab 3G3, 0.5 mg/kg xisomab 3G3, or matching placebo on Day 1 at Hour 0. The dose will be administered proximal to the dialyzer cartridge, into the arterial line immediately after start of HD.

Planned doses for each cohort of the study are as follows:

Cohort 1: 0.25 mg/kg xisomab 3G3 or matching placebo Cohort 2: 0.5 mg/kg xisomab 3G3 or matching placebo

The patients' weight recorded at check-in will be used to calculate the study drug dose.

Treatments will be described as follows:

| Cohort | Treatment | Short Description (used in text) | Long Description (used in<br>Tables Figures and Listings) |
|---|---|---|---|
| Cohorts 1 & 2 | P | Placebo (Pooled) | Single IV Infusion of Placebo (Pooled) |
| Cohort 1 | A | 0.25 mg/kg<br>xisomab 3G3 | Single IV Infusion of 0.25 mg/kg xisomab 3G3 |
| Cohort 2 | В | 0.5 mg/kg<br>xisomab 3G3 | Single IV Infusion of 0.5 mg/kg xisomab 3G3 |

#### 6. PHARMACOKINETIC ANALYSIS

#### 6.1 Measurements and Collection Schedule

For all patients, blood samples for the determination of free xisomab 3G3 will be collected at predose (hour 0, at least 1 hour prior the start of HD session) and at 0.167, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 96, 120, 144, and 192 hours after xisomab 3G3 start of infusion.

All concentration data will be included in the calculation of the individual PK parameters, the individual concentration-time plots (based on actual sample times), and in the mean concentration-time plots (based on nominal sample times). However, if there are any significant deviations from nominal sample times, some concentration data may be excluded from mean concentration-time plots and/or additional concentration-time plots of the mean data may be provided. All deviations and excluded data will be provided and discussed in the CSR.

## 6.2 Bioanalytical Method

Plasma concentrations of xisomab 3G3 will be determined using enzyme-linked immunosorbent assay (ELISA) validated with respect to accuracy, precision,

linearity, sensitivity, and specificity at Celerion, Lincoln, Nebraska. The analytical range (lower limit of quantitation [LLOQ] – upper limit of quantitation [ULOQ]) for xisomab 3G3 is expected to be 50 – 5000 ng/mL.

### 6.3 Investigational Product and PK Analyte Information

#### **6.3.1** Xisomab 3G3

Xisomab 3G3 is a novel, injectable, therapeutic monoclonal antibody (IgG4, S241P hinge-modified) that prevents activation of the contact (intrinsic) pathway of coagulation and is intended to address the problem of dose limiting bleeding side effects of current antithrombotic agents. Xisomab 3G3 was developed by Aronora, Inc. and is intended for IV administration. The proposed indication for xisomab 3G3 is as a therapeutic treatment of venous thromboembolism. The goal of xisomab 3G3 treatment is to achieve safe anticoagulation for several days with a single dose.

Xisomab 3G3 and matching placebo was supplied as sterile powder for injection via the IV route, upon reconstitution.

The quantity referenced for doses are based on active drug substance (i.e., xisomab 3G3); therefore, dose adjustment is not required for calculation of dose-dependent PK parameters for the parent drug.

#### 6.4 Pharmacokinetic Concentrations

Plasma concentrations of xisomab 3G3 as determined at the collection times and per the bioanalytical method described in Section 6.1 and Section 6.2, respectively, will be used for the calculation of the plasma xisomab 3G3 PK parameters.

#### 6.5 Noncompartmental Pharmacokinetic Analysis and Parameter Calculation

#### 6.5.1 Plasma Pharmacokinetic Parameters

The appropriate noncompartmental PK parameters will be calculated from the plasma free xisomab 3G3 concentration-time data using Phoenix® WinNonlin® Version 7.0 or higher. Actual sample times will be used in the calculations of the PK parameters. The calculation of the actual time for xisomab 3G3 will be in respect to the start of infusion time of xisomab 3G3 on Day 1. All PK parameters included in the protocol are listed in Table 6.1 below, and are defined as appropriate for study design.

Table 6.1. Noncompartmental Pharmacokinetic Parameters to be Calculated

| Parameter<br>Label to be<br>Used in the | | |
|---|---|---|
| Text, Tables and Figures | Definition | Method of Determination |
| AUC0-t | Area under the concentration-time curve from time 0 to the time of the last measurable non-zero concentration | Calculated using the Linear<br>Trapezoidal with Linear<br>Interpolation Method |
| AUC0-inf | Area under the concentration-time curve from time 0 extrapolated to infinity | AUC0-inf = AUC0-t + (Clast/kel) where Clast is the last observed/measured concentration |
| AUC%extrap | Percent of AUC0-inf extrapolated | AUC%extrap =<br>(1 - AUC0-t/AUC0-<br>inf)*100 |
| AUMC0-inf* | Area under the moment curve from time 0 extrapolated to infinity | AUMC0-inf = AUMC0-t + [(tlast x Clast)/ Kel]+<br>[Clast/(Kel) <sup>2</sup> ] |
| Cmax | The maximum observed concentration | Taken directly from bioanalytical data |
| Tmax | The time to reach Cmax. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value | Taken from clinical database as the difference in the start time of the infusion and the time of the blood draw which is associated with the Cmax. |
| Kel | Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma concentration versus time curve | The parameter will be calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase (e.g., three or more non-zero plasma concentrations). |
| t½ | Apparent first-order terminal elimination half-life | Calculated as: 0.693/ Kel |
| CL | The apparent total plasma clearance after IV administration | Calculated as:<br>Dose/(AUC0-inf) |
| MRT* | Mean residence time of free drug in the systemic circulation when the drug concentrations are extrapolated to infinity | Calculated as:<br>(AUMC0-inf/AUC0-inf) –<br>(T1/2)<br>Where TI is the duration of<br>infusion |
| Vss | Total apparent volume of distribution following single IV dose administration | Calculated as:<br>MRT x CL |

\* AUMC0-inf and MRT values will be used for Vss calculation but will not be listed in the PK tables. Note for the programmer: Parameters which are calculated for use in the calculation of a separate parameter but that are not summarized in the PK tables (i.e., AUMC0-inf and MRT) will be included in the study data tabulation model (SDTM) PP(Pharmacokinetic Parameters) domain, but not included in the analysis data model (ADaM) ADPP (Pharmacokinetic Parameters Analysis) domain.

PK parameters will not be calculated for patients with 2 or fewer consecutive time points with detectable concentrations. Subjects for whom there are insufficient data to calculate the PK parameters will be included in the concentration tables only and excluded from the summary statistics.

For the calculation of the PK parameters, plasma concentrations below the limit of quantitation (BLQ) prior to the first quantifiable concentration will be set to 0 and plasma concentrations BLQ after the first quantifiable concentration will be treated as missing.

The Kel will be determined using linear regressions composed of least 3 data points. The Kel will not be assigned if 1) the terminal elimination phase is not apparent, 2) if Tmax is one of the 3 last data points, or 3) if the R<sup>2</sup> value is less than 0.75. In cases where the Kel interval is not assigned, the values of AUC0-inf, AUC%extrap, AUMC0-inf, t½, CL, MRT, and Vss are considered not calculable and will not be reported. Wherever the resulting t½ is more than half as long as the sampling interval, the Kel values and associated parameters (AUC0-inf, AUC%extrap, AUMC0-inf, t½, CL, MRT, and Vss) may not be presented as judged appropriate and in accordance with Celerion SOPs.

#### 6.6 Data Summarization and Presentation of PK Parameters

All plasma xisomab 3G3 PK concentrations and/or PK parameters descriptive statistics will be generated using SAS® version 9.3 or higher. A concentration table will be presented for pooled placebo samples without descriptive statistics.

The plasma concentrations of xisomab 3G3 will be listed and summarized by treatment and time points for all subjects in the PK population. Plasma concentrations of xisomab 3G3 will be presented with the same level of precision as received from the bioanalytical laboratory. Summary statistics, including sample size (n), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV%), standard error of the mean (SEM), minimum, median, and maximum will be calculated for all nominal concentration time points. Excluded subjects will be included in the concentration listings, but will be excluded from the summary statistics and noted as such in the tables. All BLQ values will be presented as "BLQ" in the concentration listings and footnoted accordingly.

Mean and individual concentration-time profiles will be presented on linear and semi-log scales. Linear mean plots will be presented with and without SD.

Plasma xisomab 3G3 PK parameters will be listed and summarized by treatment for all subjects in the PK population. Pharmacokinetic parameters will be reported to 3 significant figures for individual parameters, with the exception of t½ and Tmax, which will be presented with 2 decimal places. Summary statistics (n, Mean, SD, CV%, SEM, minimum, median, maximum, geometric mean [Geom Mean] and geometric CV% [Geom CV%]) will be calculated for plasma xisomab 3G3 PK parameters. Excluded subjects will be listed in the PK parameter tables, but will be excluded from the summary statistics and noted as such in the tables.

The level of precision for each concentration and PK parameter statistic will be presented as follows:

- minimum/maximum: in same precision as in the bioanalytical data for concentrations and same precision for PK parameters presentation
- Mean/median/Geom Mean: in one more level of precision than minimum/maximum
- SD/SEM: in one more level of precision than Mean/median/Geom Mean
- n will be presented as an integer
- CV% and Geom CV% will be presented to the nearest tenth

#### 7. PHARMACODYNAMICS

## 7.1 Pharmacodynamic Assessment

Pharmacodynamic (PD) assessment will include evaluation of drug potency and efficiency of HD.

#### 7.1.1 Drug potency

Drug potency will be evaluated using the following PD markers:

- Thrombus accumulation will be evaluated by a visual inspection of the dialyzer membrane at the end of HD procedures and by a gradation using a standardized visual assessment scale;
- Total protein accumulation within the HD filter will be evaluated using appropriate methods;
- Coagulation parameter (activated partial thromboplastin time [aPTT]).

#### 7.1.2 Efficiency of HD

Efficiency of HD will be assessed by:

- Blood BUN and potassium levels before and after dialysis;
- Length of HD will be calculated as end time minus start time in hours and presented in individual and mean tables for each treatment;

- Total dialysate urea (measurement of BUN removed over 4 hours of dialysis) will be used to calculate;
  - o Single pool Kt/V. The formula to calculate Kt/V is listed under Section 7.2.3.
  - URR measured as the difference between urea pre-dialysis and post-dialysis expressed as a percentage. The formula to calculate URR is listed under Section 7.2.3.

#### 7.2 Data Summarization and Presentation of PD Parameters

#### 7.2.1 aPTT

Sample Collection: Samples for the coagulation parameter (aPTT) will be collected at screening, pre- and post-dialysis on Days -7, -5, -3, 1, 3, 5, and 12. Additional samples for aPTT will be collected following xisomab 3G3/placebo dosing on Day 1 at predose (hour 0, at least 1 hour prior the start of HD session) and at 0.167, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 96, 120, 144, and 192, hours after xisomab 3G3 start of infusion.

**Baseline Calculation Method Following Day 1 Dosing:** Following xisomab 3G3 dosing on Day 1, aPTT change from baseline will be calculated by dividing postdose aPTT values from average of pre-dose baseline (the average of pre-dialysis aPTT values on Days -7, -5, -3, and 1 will be calculated as pre-dose baseline).

<u>Fold change in aPTT values:</u> The fold change in aPTT values on Days -7, -5, -3, 1 (only pre- and post-dialysis aPTT values on Day 1), 3, 5, and 12 will be calculated by dividing the post-dialysis aPTT/pre-dialysis aPTT values for each day separately.

aPTT values will be extracted from the clinical laboratory database and descriptive statistics will be generated using SAS® version 9.3 or higher. Following Day 1 xisomab 3G3 dosing, a table will be presented for the aPTT change from baseline with descriptive statistics.

aPTT values will be listed and summarized by treatment and time points in Tables and Figures for all subjects in the Safety Population (2 active dose levels and pooled placebo). aPTT values will be presented with the same level of precision as received from the clinical laboratory database. Summary statistics, including n, Mean, SD, CV%, SEM, minimum, median, and maximum will be calculated for all nominal values time points. Excluded subjects will be included in the aPPT values tables, but will be excluded from the summary statistics and noted as such in the tables.

Mean and individual aPTT values-time and change from baseline-time profiles will be presented on linear scale. Linear mean plots will be presented with and without SD.

The level of precision for the aPPT values summary statistic will be presented as follows:

- minimum/maximum: in same precision as in the clinical laboratory database
- Mean/median: in one more level of precision than minimum/maximum
- SD/SEM: in one more level of precision than Mean/median
- n will be presented as an integer
- CV% will be presented to the nearest tenth

#### 7.2.2 BUN and Potassium:

Sample Collection: Samples for BUN and potassium will be collected pre- and post-dialysis on Days -7, -5, -3, 1, 3, 5, and 12.

Change in BUN and Potassium values: The change in BUN values on Days -7, -5, -3, 1, 3, 5, and 12 will be calculated by subtracting the post-dialysis BUN from the pre-dialysis BUN values for each day separately. The same method will be used for potassium.

Potassium and BUN values will be listed and summarized by treatment and Day in Tables and Figures for all subjects in the Safety Population (2 active dose levels and pooled placebo).

The level of precision for potassium and BUN summary statistic will be the same as per aPTT values listed in Section 7.2.1.

#### 7.2.3 URR and KT/V

The derived PD parameters (URR and KT/V) will be calculated from the pre- and post-dialysis BUN values on Days -7, -5, 1, 3, 5, and 12.

URR will be calculated using the following formula:

Kt/V will be calculated using the following formula:

$$sp\frac{Kt}{V} = \ln(R - (0.008 \times t)) + (4 - (3.5 \times R)) \times \frac{UF}{Wt}$$

Where R = BUN Post-dialysis/BUN Pre-dialysis

t = Time of HD

UF = Pre-dialysis Weight – Post-dialysis Weight

Wt = Post-dialysis weight of patient.

URR and Kt/V values will be listed and summarized by treatment and Day in Tables for all subjects in the Safety Population (2 active dose levels and pooled placebo).

The level of precision for URR and Kt/V summary statistic will be the same as per aPTT values listed in Section 7.2.1

### 7.2.4 Clotting in the Drip Chamber and Dialysis Filter

Visual inspection of clotting in the drip chamber will be recorded 2 hours after start of dialysis and at the end of dialysis on Days -7, -5, -3, 1, 3, 5, and 12.

Visual inspection of clotting in the dialysis filter will be recorded at the end of dialysis on Days -7, -5, -3, 1, 3, 5, and 12.

Summary of clotting values will be listed and summarized by treatment and Day in Tables for all subjects in the Safety Population (2 active dose levels and pooled placebo).

## 7.2.5 Dialysate Analysis

A 10 mL dialysate sample will be taken at the start and at the end of HD on Days -7, -5, 3, 12 and at 0.5 and 4 hours post dosing on Day 1.

The samples will be sent to Aronora and will be stored for up to 5 years following the last dosing for future analysis (e.g., xisomab 3G3 levels and or urea).

#### 8. SAFETY

All case report form (CRF) data will be listed by subject and chronologically by assessment time points. This will include rechecks, unscheduled assessments, and early termination.

Applicable continuous variables will be summarized using n, arithmetic mean, SD, minimum, median, and maximum. Data from subjects who received the placebo treatment will be pooled across cohorts.

The level of precision will be presented as follows: minimum/maximum in the same precision as in the database, mean/median in one more precision level than minimum/maximum, SD in one more precision level than mean/median, and n will be presented as an integer. Percentages of total frequency counts, if presented, will be reported as whole numbers.

Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators.

#### 8.1 Subject Discontinuation

Subjects will be summarized by number of subjects dosed, completed, and discontinued the study with discontinuation reasons by treatment (two dose levels and pooled placebo and study overall.

## 8.2 Demographics

Descriptive statistics will be calculated for continuous variables (age, weight, height, and body mass index) and frequency counts will be provided for categorical variables (race, ethnicity, and sex) by treatment and overall. Age will be derived from date of birth to date of first dosing.

#### **8.3** Adverse Events

All adverse events (AEs) occurring during this clinical trial will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®), Version 21.1.

All AEs captured in the database will be listed in by-subject data listings including verbatim term, coded term, treatment, severity, relationship to study medication, and action; however, only treatment-emergent AEs (TEAEs) will be summarized.

A TEAE is defined as an AE that is starting or worsening at the time of or after study drug administration. Each TEAE will be attributed to a treatment based on the onset date and time of the AE. If the onset time of an AE is missing and the onset date is the same as the treatment dosing date, then the AE will be considered treatment emergent. If the onset date of an AE is missing, then the AE will be considered treatment emergent.

TEAEs will be tabulated by System Organ Class (SOC) and Preferred Term. Summary tables will include number of subjects reporting the AE and as percent of number of subjects dosed by treatment and overall. The number of AEs will be tabulated in a similar manner. Tables which tabulate the number of TEAEs by severity and relationship to study treatment will also be included.

Serious adverse events (SAEs), if present, will also be listed. Applicable narratives will be included in the CSR.

## 8.4 Clinical Laboratory Tests (Serum Chemistry, Hematology, Coagulation and Urinalysis)

Safety serum chemistry, hematology and urinalysis tests are performed at Screening, Day -8 check-in, Day 1 predose, Day 6 and Day 12. For anuric patients, urinalysis may not be performed. Platelet count are collected at start and end of HD on Days -7, -5, -3, 1, 3, 5 and 12 and on Day 6. Platelet count are collected at start and end of HD on Days -7, -5, -3, 1, 3, 5 and 12 and Day 6. aPTT results are presented and discussed in the PD Section 7.2.

Out-of-range values and clinically significant results will be listed.

For all numeric laboratory values, descriptive statistics will be presented for each laboratory test by assessment time point and treatment. Change from baseline will be summarized in a similar manner. Baseline is defined as the result closest and prior to

dose which may include unscheduled results. This will typically be the result collected at predose on Day 1. Postdose unscheduled events or early termination results will not be included in summaries.

For each laboratory test, a shift table will be developed to compare the frequency of the results at baseline (above normal, normal, or below normal) with the respective postdose results.

Coagulation parameters and platelet count will be listed and presented together since they have the same timepoints. Urinalysis test results will be listed only.

## 8.5 Vital Signs

Vital signs tests (HR, BP, RR and T) will be assessed at Screening, Day -8 check-in, start of HD on Days -7, -5, -3, 1, 3, 5, 8, 10 and 12, 1 hour postdose on Day1, Day 6 discharge or early term and Day 12 follow-up.

Vital sign results will be summarized by dose level, pooled placebo, and time point. Change from baseline will be summarized in a similar way. Baseline is defined as the result closest and prior to the dose on Day 1, which may include unscheduled results, whichever is later. Postdose unscheduled events or early termination results will not be included in summaries.

### 8.6 Electrocardiogram

Safety ECGs (HR, PR, QRS, QT and Fridericia correction QTcF) will be assessed at Screening, Day -8 check-in, Day 1 predose, Day 6 (discharge or early term) and Day 12 follow-up.

ECG parameters will be summarized by dose level, pooled placebo, and time point. Change from baseline will be summarized in a similar way. Baseline is defined as the result closest and prior to the dose on Day 1, which may include unscheduled results, whichever is later. Postdose unscheduled events or early termination results will not be included in summaries.

The QTcF values that are > 450 ms and increase from baseline > 30 ms, will be flagged in the data listings.

#### 8.7 Concomitant Medications

All concomitant medications recorded during the study will be coded with the WHO Dictionary Version September 2018, B3 and listed.

#### 8.8 Physical Examination

Full physical examinations will be performed at Screening and Day -8 check-in and abbreviated physical examination will be performed on Days 1, 6 and 12. Abnormal findings will be reported as medical history or adverse events. All data found in the CRF will be listed.

#### **8.9** Vascular Access Site Reaction

Vascular access site reaction will be assessed at predose on Day 1 and end of HD on Days 1, 3 and 5. Any new abnormal findings inconsistent with past skin injuries as expected in patient on chronic HD will be reported as AEs.

#### **8.10** Bleeding Time

The time to clot (bleeding time) will be recorded following hemodialysis after the needle is removed from the vascular access site on Days -7, -5, -3, 1, 3, 5 and 12. Summary statistics will be calculated for time to clot by treatment and assessment timepoint.

### 8.11 Medical History

All medical and surgical histories recorded in the study will be coded with MedDRA®, Version 21.1. and listed.

## 8.12 Immunogenecity

Development of antibodies against the study drug will be evaluated by determining the anti-drug antibody (ADA) titer.

Blood samples will be collected from each subject for ADA detection prior to dosing on Day 1 and at the end of HD on Day 12. Immunogenicity testing will be done at Celerion, Lincoln, Nebraska.

Summary counts of positive and negative ADA detection will be presented by collection time and treatment.

#### 9. SUMMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS

The length of HD was 3 hours in the protocol and should be approximately 4 hours. The samples collected for BUN and potassium will be at the end of dialysis (approximately 4 hours).

The analyses described in this SAP are aligned with those analyses described in the protocol.

#### 10. SUMMARY TABLES AND FIGURES

Summary tables and figures are numbered following the International Conference on Harmonization (ICH) structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. Note that all PK, PD, immunogenicity and Safety summary tables and figures will be generated using SAS®

Version 9.3 or higher and/or using Phoenix® WinNonlin® Version 7.0 or higher for summary PK TFLs, as appropriate.

## 10.1 In-text Summary Tables and Figures

The following is a list of table and figure titles that will be included in the text of the CSR. Tables and figures will be numbered appropriately during compilation of the CSR.

## Section 10:

Table 10-1 Subject Disposition Summary

#### Section 11:

- Table 11-1 Demographic Summary
- Table 11-2 Summary of Plasma Xisomab 3G3 Pharmacokinetics Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 (Pharmacokinetic Population)

#### **Efficiency of HD:**

- Table 11-3 Summary of Difference Between Pre- and Post-dialysis BUN and URR Days -7 to 12 (Safety Population)
- Table 11-4 Summary of Difference Between Pre- and Post-dialysis Potassium Days -7 toSummary 12 (Safety Population)
- Table 11-5 Summary of Kt/V Values (Safety Population)

#### **Drug Potency:**

- Table 11-6 Summary of Difference Between Pre- and Post-dialysis aPTT Days -7 to 12 (Safety Population)
- Table 11-7 Summary of Clotting in the Drip Chamber Days -7 to 12 (Safety Population)
- Table 11-8 Summary of Clotting in the Dialysis Filter Days -7 to 12 (Safety Population)

#### **Figures**

- Figure 11-1 Arithmetic Mean Plasma Xisomab 3G3 Concentration Versus Time Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 (Linear Scale) (Pharmacokinetic Population)
- Figure 11-2 Arithmetic Mean Pre- and Post-dialysis BUN Values Days -7 to 12 (Linear Scale) (Safety Population)
- Figure 11-3 Arithmetic Mean Pre- and Post-dialysis Potassium Values Days -7 to 12 (Linear Scale) (Safety Population)

| Figure 11-4 | Arithmetic Mean aPPT Values Versus Time Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 and Placebo (Pooled) – Day 1 (Linear Scale) (Safety Population) |
|---|---|
| Figure 11-5 | Arithmetic Mean aPPT Values Versus Time During the Course of the Study – Days -7 to 12 (Linear Scale) (Safety Population) |
| Figure 11-6 | Arithmetic Mean aPPT Change From Baseline Versus Time Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 and Placebo (Pooled) – Day 1 (Linear Scale) (Safety Population) |
| Figure 11-7 | Arithmetic Mean pre- and Post-dialysis aPTT Values – Days -7 to 12 (Linear Scale) (Safety Population) |
| Section 12: | |
| Table 12-1 | Adverse Event Frequency by Treatment - Number of Subjects<br>Reporting the Event (% of Subjects Dosed) |
| Table 12-2 | Summary of Difference Between Pre- and Post-dialysis PT – Days -7 to 12 (Safety Population) |
| Table 12-3 | Summary of Difference Between Pre- and Post-dialysis INR – Days -7 to 12 (Safety Population) |
| Table 12-4 | Summary of Difference Between Pre- and Post-dialysis PT/INR – Days -7 to 12 (Safety Population) |
| Table 12-5 | Summary of Post-dialysis Bleeding Time – Days -7 to 12 (Safety |

#### **10.2** Section 14 Summary Tables and Figures

Population)

The following is a list of table and figure titles that will be included in Section 14 of the report. Table and figure titles may be re-numbered as appropriate during the compilation of the report.

#### 14.1 Demographic Data Summary Tables

The following is a list of table and figure titles that will be included in Section 14 of the report. Table and figure titles may be renumbered as appropriate during the compilation of the report.

- Table 14.1.1 Summary of Disposition (Safety Population)
- Table 14.1.2 Summary of Demographics (Safety Population)

## 14.2 Pharmacokinetic and Pharmacodynamic Data Summary Tables and Figures

## **Pharmacokinetic Tables and Figures**

#### 14.2.1. Plasma Pharmacokinetic Xisomab 3G3 Tables and Figures

- Table 14.2.1.1.1 Plasma Xisomab 3G3 Concentrations (ng/mL) Following a Single IV Infusion of 0.25 mg/kg Xisomab 3G3 (Pharmacokinetic Population)
- Table 14.2.1.1.2 Plasma Xisomab 3G3 Concentrations (ng/mL) Following a Single IV Infusion of 0.5 mg/kg Xisomab 3G3 (Pharmacokinetic Population)
- Table 14.2.1.1.3 Plasma Xisomab 3G3 Concentrations (ng/mL) Following a Single IV Infusion of Placebo (Pooled)
- Table 14.2.1.1.4 Plasma Xisomab 3G3 Pharmacokinetic Parameters Following a Single IV Infusion of 0.25 mg/kg Xisomab 3G3 (Pharmacokinetic Population)
- Table 14.2.1.1.5 Plasma Xisomab 3G3 Pharmacokinetic Parameters
  Following a Single IV Infusion of 0.5 mg/kg Xisomab 3G3
  (Pharmacokinetic Population)
- Table 14.2.1.1.6 Intervals (Hours) Used for Determination of Plasma Xisomab 3G3 Kel Values (Pharmacokinetic Population)
- Figure 14.2.1.2.1 Arithmetic Mean (SD) Plasma Xisomab 3G3 Concentration Versus Time Profiles Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 (Linear Scale) (Pharmacokinetic Population)
- Figure 14.2.1.2.2 Arithmetic Mean Plasma Xisomab 3G3 Concentration Versus Time Profiles Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 (Linear Scale) (Pharmacokinetic Population)
- Figure 14.2.1.2.3 Arithmetic Mean Plasma Xisomab 3G3 Concentration Versus Time Profiles Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 (Semi-Log Scale) (Pharmacokinetic Population)

## Pharmacodynamic/Immunogenicity Tables and Figures

#### 14.2.2 BUN Tables and Figures

- Table 14.2.2.1.1 Individual and Mean Difference Between Pre- and Post-dialysis BUN Values (unit) and URR Days -7 to 12 0.25 mg/kg Xisomab 3G3 on Day 1 (Safety Population)
- Table 14.2.2.1.2 Individual and Mean Difference Between Pre- and Postdialysis BUN Values (unit) and URR – Days -7 to 12 – 0.5 mg/kg Xisomab 3G3 on Day 1 (Safety Population)

Table 14.2.2.1.3 Individual and Mean Difference Between Pre- and Postdialysis BUN Values (unit) and URR – Days -7 to 12 – Placebo (Pooled) (Safety Population)

#### **Programmer Note:**

For Tables 14.2.2.1.1 through 14.2.2.1.3, the difference will be calculated as follows: (Pre-dialysis – Post-dialysis).

- Figure 14.2.2.2.1 Arithmetic Mean Pre- and Post-dialysis BUN Values Days -7 to 12 (Linear Scale) (Safety Population)
- Figure 14.2.2.2.2 Arithmetic Mean (SD) Pre- and Post-dialysis BUN Values Days -7 to 12 (Linear Scale) (Safety Population)

## **14.2.3** Potassium Tables and Figures

- Table 14.2.3.1.1 Individual and Mean Difference Between Pre- and Postdialysis Potassium Values (unit) – Days -7 to 12 – 0.25 mg/kg Xisomab 3G3 on Day 1 (Safety Population)
- Table 14.2.3.1.2 Individual and Mean Difference Between Pre- and Post-dialysis Potassium Values (unit) Days -7 to 12 0.5 mg/kg Xisomab 3G3 on Day 1 (Safety Population)
- Table 14.2.3.1.3 Individual and Mean Difference Between Pre- and Postdialysis Potassium Values (unit) – Days -7 to 12 – Placebo (Pooled) (Safety Population)

## <u>Programmer Note:</u>

For Tables 14.2.3.1.1 through 14.2.3.1.3, the difference will be calculated as follows: (Pre-dialysis – Post-dialysis).

- Figure 14.2.3.2.1 Arithmetic Mean Pre- and Post-dialysis Potassium Values Days -7 to 12 (Linear Scale) (Safety Population)
- Figure 14.2.3.2.2 Arithmetic Mean (SD) Pre- and Post-dialysis Potassium Values Days -7 to 12 (Linear Scale) (Safety Population)

#### **14.2.4** Kt/V Tables

- Table 14.2.4.1.1 Individual and Mean Kt/V Values (unit) 0.25 mg/kg Xisomab 3G3 on Day 1 (Safety Population)
- Table 14.2.4.1.2 Individual and Mean Kt/V Values (unit) 0.5 mg/kg Xisomab 3G3 on Day 1 (Safety Population)
- Table 14.2.4.1.3 Individual and Mean Kt/V Values (unit) Placebo (Pooled) (Safety Population)

#### 14.2.5 aPTT Tables and Figures

Table 14.2.5.1.1 Individual and Mean aPTT Values (unit) During the Course of the Study (Days -7 to 12) and Following a Single IV

| Table 14.2.5.1.2 | Infusion of 0.25 mg/kg Xisomab 3G3 on Day 1 (Safety Population) Individual and Mean aPTT Values (unit) During the Course of the Study (Days -7 to 12) and Following a Single IV Infusion of 0.5 mg/kg Xisomab 3G3 on Day 1 (Safety |
|---|---|
| Table 14.2.5.1.3 | Population) Individual and Mean aPTT Values (unit) During the Course of the Study (Days -7 to 12) and Following a Single IV Infusion of Placebo (Pooled) on Day 1 (Safety Population) |
| Table 14.2.5.1.4 | Individual and Mean aPTT Change From Baseline Values (unit) Following a Single IV Infusion of 0.25 mg/kg Xisomab 3G3 on Day 1 (Safety Population) |
| Table 14.2.5.1.5 | Individual and Mean aPTT Change From Baseline Values (unit) Following a Single IV Infusion of 0.5 mg/kg Xisomab 3G3 on Day 1 (Safety Population) |
| Table 14.2.5.1.6 | Individual and Mean aPTT Change From Baseline Values (unit) Following a Single IV Infusion of Placebo (Pooled) – Day 1 (Safety Population) |
| <u>Programmer Note:</u> | For Tables 14.2.5.1.4 through 14.2.5.1.6, aPTT baseline will be the average of all pre-dialysis aPTT value on |
| | Days -7, -5, -3 and 1, and the change from baseline will be calculated as follows: (post-dialysis/baseline). |
| Table 14.2.5.1.7 | <i>calculated as follows: (post-dialysis/baseline).</i> Individual and Mean Difference Between Pre- and Post-dialysis aPTT Values (unit) – Days -7 to 12 – 0.25 mg/kg |
| Table 14.2.5.1.7 Table 14.2.5.1.8 | calculated as follows: (post-dialysis/baseline). Individual and Mean Difference Between Pre- and Post- |
| | Individual and Mean Difference Between Pre- and Post-dialysis aPTT Values (unit) – Days -7 to 12 – 0.25 mg/kg Xisomab 3G3 on Day 1 (Safety Population) Individual and Mean Difference Between Pre- and Post-dialysis aPTT Values (unit) – Days -7 to 12 – 0.5 mg/kg |
| Table 14.2.5.1.8 | Individual and Mean Difference Between Pre- and Post-dialysis aPTT Values (unit) – Days -7 to 12 – 0.25 mg/kg Xisomab 3G3 on Day 1 (Safety Population) Individual and Mean Difference Between Pre- and Post-dialysis aPTT Values (unit) – Days -7 to 12 – 0.5 mg/kg Xisomab 3G3 on Day 1 (Safety Population) Individual and Mean Difference Between Pre- and Post-dialysis aPTT Values (unit) – Days -7 to 12 – Placebo |

- Figure 14.2.5.2.2 Arithmetic Mean (SD) aPPT Values Versus Time Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 and Placebo (Pooled) Day 1 (Linear Scale) (Safety Population)
- Figure 14.2.5.2.3 Arithmetic Mean aPPT Values Versus Time During the Course of the Study Days -7 to 12 (Linear Scale) (Safety Population)
- Figure 14.2.5.2.4 Arithmetic Mean (SD) aPPT Values Versus Time During the Course of the Study Days -7 to 12 (Linear Scale) (Safety Population)
- Figure 14.2.5.2.5 Arithmetic Mean aPPT Change From Baseline Versus Time Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 and Placebo (Pooled) Day 1 (Linear Scale) (Safety Population)
- Figure 14.2.5.2.6 Arithmetic Mean (SD) aPPT Change From Baseline Versus
  Time Following a Single IV Infusion of 0.25 and 0.5 mg/kg
  Xisomab 3G3 and Placebo (Pooled) Day 1 (Linear Scale)
  (Safety Population)
- Figure 14.2.5.2.7 Arithmetic Mean Pre- and Post-dialysis aPTT Values Days -7 to 12 (Linear Scale) (Safety Population)
- Figure 14.2.5.2.8 Arithmetic Mean (SD) Pre- and Post-dialysis aPTT Values Days -7 to 12 (Linear Scale) (Safety Population)

## 14.2.6 Clotting in the Drip Chamber Tables

Table 14.2.6.1 Summary of Clotting in the Drip Chamber (Safety Population)

## 14.2.7 Clotting in Dialysis Filter Tables

Table 14.2.7.1 Summary of Clotting in the Dialysis Filter (Safety Population)

#### 14.3 Safety Data Summary Tables

## 14.3.1 Displays of Adverse Events

Table 14.3.1.1 Treatment-emergent Adverse Event Frequency by Treatment

- Number of Subjects Reporting the Event (% of Subject Dosed) (Safety Population)

- Table 14.3.1.2 Treatment-emergent Adverse Event Frequency by Treatment

   Number of Adverse Events (% of Total Adverse Events)

  (Safety Population)
- Table 14.3.1.3 Treatment-emergent Adverse Event Frequency by Treatment, Severity, and Relationship to Drug Number of Adverse Events (Safety Population)

#### 14.3.2 Listings of Deaths, other Serious and Significant Adverse Events

Table 14.3.2.1 Serious Adverse Events (Safety Population)

<if no serious adverse event occurred, a statement 'No serious adverse event is reported'>

## 14.3.3 Narratives of Deaths, other Serious and Certain other Significant Adverse Events

#### 14.3.4 Abnormal Laboratory Value Listing (each patient)

- Table 14.3.4.1 Out-of-Range Values and Recheck Results Serum Chemistry (Safety Population)
- Table 14.3.4.2 Out-of-Range Values and Recheck Results Hematology/Coagulation (Safety Population)
- Table 14.3.4.3 Out-of-Range Values and Recheck Results Urinalysis (Safety Population)

## 14.3.5 Displays of Other Laboratory, Vital Signs, Electrocardiogram, Physical Examination, and Other Safety Data

- Table 14.3.5.1 Clinical Laboratory Summary and Change from Baseline Serum Chemistry (Safety Population)
- Table 14.3.5.2 Clinical Laboratory Shift from Baseline Serum Chemistry (Safety Population)
- Table 14.3.5.3 Clinical Laboratory Summary and Change from Baseline Hematology (Safety Population)
- Table 14.3.5.4 Clinical Laboratory Shift from Baseline Hematology (Safety Population)
- Table 14.3.5.5 Clinical Laboratory Summary and Change from Baseline Coagulation and Platelet Count (Safety Population)
- Table 14.3.5.6 Clinical Laboratory Shift from Baseline Coagulation and Platelet Count (Safety Population)
- Table 14.3.5.7 Vital Sign Summary and Change from Baseline (Safety Population)

Table 14.3.5.8 12-Lead Electrocardiogram Summary and Change from Baseline (Safety Population)

Table 14.3.5.9 Frequency of Immunogenicity - ADA Titer (Safety Population)

#### 10.3 Section 16 Data Listings

Data listings are numbered following the ICH structure but may be renumbered as appropriate during the compilation of the TFLs for the CSR. The following is a list of appendix numbers and titles that will be included as data listings:

## **16.1** Study Information

Appendix 16.1.9 Statistical Methods

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

### 16.2 Subject Data Listings

#### **16.2.1** Subject Discontinuation

Appendix 16.2.1 Study Completion/Early Termination (Safety Population)

#### **16.2.2** Protocol Deviations

Appendix 16.2.2 Protocol Deviations

## 16.2.3 Subjects Excluded from Pharmacokinetic/Pharmcodynamic Analyses

Appendix 16.2.3 Subjects Excluded from Pharmacokinetic/Pharmacodynamic Analyses

<Note: Appendices 16.2.2 and 16.2.3 are generated in MS Word for inclusion in the study report.>

## 16.2.4 Demographic Data

| Appendix 16.2.4.1 | Demographics (Safety Population) |
|-------------------|--------------------------------------------------|
| Appendix 16.2.4.2 | Physical Examination (Safety Population) |
| Appendix 16.2.4.3 | Medical and Surgical History (Safety Population) |
| Appendix 16.2.4.4 | Alcohol Screen (Safety Population) |
| Appendix 16.2.4.5 | Drug Screen (Safety Population) |

#### 16.2.5 Compliance and/or Drug Concentration Data

| Appendix 16.2.5.1 | Subject Eligibility (Safety Population) |
|---|---|
| Appendix 16.2.5.2 | Subject Eligibility at Check-In (Safety Population) |
| Appendix 16.2.5.3 | Test Compound Administration (Safety Population) |
| Appendix 16.2.5.4 | Blood Draw Times for Free xisomab 3G3 PK (Safety Population) |
| Appendix 16.2.5.5 | Blood Draw Times for Free xisomab 3G3 PD (aPTT) (Safety Population) |
| Appendix 16.2.5.6 | Blood Draw Times for Immunogenicity (Safety Population) |
| Appendix 16.2.5.7 | Blood Draw Times for Dialysate Analysis for Kt/V and URR (Safety Population) |
| Appendix 16.2.5.8.1 | Dialyzer Assessment (I of V) (Safety Population) |
| Appendix 16.2.5.8.2 | Dialyzer Assessment (II of V) (Safety Population) |
| Appendix 16.2.5.8.3 | Dialyzer Assessment (III of V) – (Safety Population<br>Number and Volume of Saline Flushes) |
| Appendix 16.2.5.8.4 | Dialyzer Assessment (IV of V) – Clotting in Drip<br>Chamber (Safety Population) |
| Appendix 16.2.5.8.5 | Dialyzer Assessment (V of V) – Clotting in Dialysis Filter (Safety Population) |
| Appendix 16.2.5.9 | Non-Study Procedures (Safety Population) |
| Appendix 16.2.5.10 | Prior and Concomitant Medications (Safety Population) |

## 16.2.6 Individual Pharmacokinetic Response Data

## **Individual Xisomab 3G3 Figures**

- Appendix 16.2.6.1.1 Individual Plasma Xisomab 3G3 Concentrations Versus Time Profiles Following a Single IV Infusion of 0.25 mg/kg Xisomab 3G3 (Linear and Semi-Log Scale) for <Subject #>
- Appendix 16.2.6.1.2 Individual Plasma Xisomab 3G3 Concentrations Versus Time Profiles Following a Single IV Infusion of 0.5 mg/kg Xisomab 3G3 (Linear and Semi-Log Scale) for <Subject #>
- Appendix 16.2.6.2.1 Individual aPTT Values Versus Time Profiles During the Course of the Study (Linear Scale) for <Subject #>

## 16.2.7 Adverse Events Listings

| Appendix 16.2.7.1.1 | Adverse Events (I of II) (Safety Population) |
|---|---|
| Appendix 16.2.7.1.2 | Adverse Events (II of II) (Safety Population) |
| Appendix 16.2.7.2 | Adverse Event Preferred Term Classification (Safety Population) |

# 16.2.8 Listings of Individual Laboratory Measurements and Other Safety Observations

| Appendix 16.2.8.1.1 | Clinical Laboratory Report - Serum Chemistry (Safety Population) |
|---|---|
| Appendix 16.2.8.1.2 | Clinical Laboratory Report - Hematology (Safety Population) |
| Appendix 16.2.8.1.3 | Clinical Laboratory Report – Coagulation and Platelet Count (Safety Population) |
| Appendix 16.2.8.1.4 | Clinical Laboratory Report - Urinalysis (Safety Population) |
| Appendix 16.2.8.1.5 | Clinical Laboratory Report – Additional Tests (Safety Population) |
| Appendix 16.2.8.1.6 | Clinical Laboratory Report - Comments (Safety Population) |
| Appendix 16.2.8.2 | Vital Signs (Safety Population) |
| Appendix 16.2.8.3 | 12-Lead Electrocardiogram (Safety Population) |
| Appendix 16.2.8.4 | Immunogenicity ADA Titer (Safety Population) |

#### 11. TABLE AND FIGURE SHELLS

The following table shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the tables that will be presented and included in the final report. Unless otherwise noted, all tables will be presented in Times New Roman font size 8. These tables will be generated of the Celerion ADaM Version 2.1 data structure.

## 11.1 In-text Summary Tables Shells

In-text Table 10-1 will be in the following format:

## **Table 10-1 Subject Disposition Summary**

Table 10-1 Subject Disposition Summary (Safety Population)

| | Dose Level of | xisomab 3G3 | Pooled | Overall |
|---------------------|---------------|-------------|----------|----------|
| Disposition | 0.25 mg/kg | 0.5 mg/kg | Placebo | |
| Dosed | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Completed | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Discontinued | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| <reason1></reason1> | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| <reason2></reason2> | X (XX%) | X (XX%) | X (XX%) | X (XX%) |

Source: Table 14.1.1

Program: /CAXXXXX/sas\_prg/stsas/intext/t\_disp.sas DDMMMYYYY HH:MM

In-text Table 11-1 will be in the following format:

**Table 11-1 Demographic Summary** 

| | Category/ | Dose Level of | f xisomab 3G3 | Pooled | |
|---|---|---|---|---|---|
| Trait | Statistics | 0.25 mg/kg | 0.5 mg/kg | Placebo | Overall |
| Sex | Male | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Female | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Race | Asian | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Black or African American | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | White | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Ethnicity | Hispanic or Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Not Hispanic or Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Age* (yrs) | n | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX |
| Weight (kg) | n | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX |

\*Age is calculated at the time of first dosing. BMI = Body mass index

Source: Table 14.1.2

Program: /CAXXXXX/sas\_prg/stsas/intexttest/t\_dem.sas DDMMMYYYY HH:MM

Programmer note: also include height and BMI

In-text Table 11-2 will be in the following format:

Table 11-2: Summary of Plasma Xisomab 3G3 Pharmacokinetics Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 (Pharmacokinetic Population)

| Pharmacokinetic<br>Parameters | Single IV Infusion of 0.25 mg/kg<br>xisomab 3G3 | Single IV Infusion of 0.5 mg/kg<br>xisomab 3G3 |
|---|---|---|
| Param1 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param2 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param3 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param4 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |

AUCs and Cmax values are presented as geometric mean and geometric CV%, when available. Tmax values are presented as median (minimum, maximum).

Other parameters are presented as arithmetic mean ( $\pm$  SD), or just mean when SD is not available. Source: Tables 14.2.1.4 through 14.2.1.5

#### Notes for Generating the Actual Table:

Presentation of Data:

- The following PK parameters will be presented in the following order and with following units: AUCO-t <ng\*hr/mL>, AUCO-inf <ng\*hr/mL>, AUC%extrap <%>, Cmax <ng/mL>, Tmax <hr>, Kel <1/hr>, t1/2 <hr>>, CL <L/hr>>, Vss <L>
- n will be presented as an integer (with no decimal);
- Summary statistics will be presented with same precision as defined in post-text shells
- Internal template ITParl

Program: /CAXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_intext\_pkparam.sas DDMMYYYY HH:MM

Table 11-3 Summary of Difference Between Pre- and Post-dialysis BUN and URR – Days -7 to 12 (Safety Population)

| | | Mean B | lood Urea Nit | rogen (Re | ference Rar | ige xx – xx | <units>) and</units> | URR (Ref | erence Ran | ge xx – xx | <%>) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Treatments | | | | | | | | | | |
| Time<br>Point | Single IV | Infusion of 3G | 0.25 mg/kg xis | Single I | | of 0.5 mg/kg x<br>G3 | isomab | Placebo (Pooled) | | | | |
| | Pre-<br>dialysis | Post-<br>dialysis | Difference | URR<br>(%) | Pre-<br>dialysis | Post-<br>dialysis | Difference | URR<br>(%) | Pre-<br>dialysis | Post-<br>dialysis | Difference | URR<br>(%) |
| | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] |
| Day -7 | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X |
| Day -5 | XXX.X <sup>a</sup> | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X |
| Day -3 | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X |
| Day 1* | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X |
| Day 3 | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X |
| Day 5 | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X |
| Day 12 | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X | XXX.X | XXX.X | XX.X | XX.X |

Difference = Pre-dialysis - Post-dialysis

URR = (1-(post-dialysis BUN/ pre-dialysis BUN))\*100

\* - Single IV infusion of 0.25, 0.5 mg/kg xisomab 3G3 or placebo was administered on Day 1

Values will be presented as arithmetic mean

Source: Tables 14.2.2.1.1 through 14.2.2.1.3

Program: /CAXXXXX/sas prg/stsas/intext/t ae.sas DDMMMYYYY HH:MM

#### Notes for Generating the Actual Table:

- n will be presented as an integer (with no decimal);
- Summary statistics will be presented with same precision as defined in post-text shells
- Internal template ITPar1, with the following changes: n will be presented in the column title with more additional columns to be created.

Program: /CAXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYY HH:MM

Program: /CAXXXXX/sas prg/pksas/adam intext pkparam.sas DDMMYYYY HH:MM

a-n = xx

Aronora, Inc. xisomab 3G3, Protocol 3G3-18-02 Celerion, Clinical Study Report No. CA23900

## Table 11-4 will be in the following format:

Table 11-4 Summary of Difference Between Pre- and Post-dialysis Potassium – Days -7 to 12 (Safety Population)

| | | | Mean | Potassium (l | Reference Rai | ıge xx − xx <uı< th=""><th>nits&gt;)</th><th></th><th></th></uı<> | nits>) | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatments | | | | | | | | |
| Time<br>Point | Single IV | / Infusion of xisomab 3G | 0 0 | Single I | V Infusion of xisomab 3G3 | ~ ~ | Placebo (Pooled) | | |
| | Pre-<br>dialysis | Post-<br>dialysis | Difference | Pre-<br>dialysis | Post-<br>dialysis | Difference | Pre-<br>dialysis | Post-<br>dialysis | Difference |
| | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] |
| Day -7 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day -5 | XXX.X | XXX.X a | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day -3 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day 1* | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day 3 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day 5 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day 6 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day 12 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |

Difference = Pre-dialysis - Post-dialysis

Values will be presented as arithmetic mean

Source: Tables 14.2.3.1.1 through 14.2.3.1.3

Program: /CAXXXXX/sas\_prg/stsas/intext/t\_ae.sas\_DDMMMYYYY\_HH:MM

#### Notes for Generating the Actual Table:

- n will be presented as an integer (with no decimal);
- · Summary statistics will be presented with same precision as defined in post-text shells
- Internal template ITPar1, with the following changes: n will be presented in the column title with additional columns to be created.

Program: /CAXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_intext\_pkparam.sas DDMMYYYY HH:MM

a-n = xx

<sup>\* -</sup> Single IV infusion of 0.25, 0.5 mg/kg xisomab 3G3 or placebo was administered on Day 1

Aronora, Inc. xisomab 3G3, Protocol 3G3-18-02 Celerion, Clinical Study Report No. CA23900

Tables 11-6, 12-2 through 12-4 will be in the following format:

Table 11-6 Summary of Difference Between Pre- and Post-dialysis aPTT – Days -7 to 12 (Safety Population)

| | | | Mea | n aPTT (Refe | rence Range xx | x - xx < units > | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatments | | | | | | | | |
| Time<br>Point | Single IV | Infusion of 0.2 xisomab 3G3 | 5 mg/kg | Single I | V Infusion of 0.<br>xisomab 3G3 | .5 mg/kg | Placebo (Pooled) | | |
| | Pre-<br>dialysis | Post-<br>dialysis | Fold<br>Change | Pre-<br>dialysis | Post-<br>dialysis | Fold<br>Change | Pre-<br>dialysis | Post-<br>dialysis | Fold<br>Change |
| | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] | (Unit)<br>[n=xx] |
| Day -7 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day -5 | XXX.X | XXX.X a | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day -3 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day 1* | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day 3 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day 5 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day 6 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| Day 12 | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |

Fold Change = Post-dialysis/Pre-dialysis

Values will be presented as arithmetic mean

Source: Tables 14.2.5.1.7 through 14.2.5.1.9

Program: /CAXXXXX/sas prg/stsas/intext/t ae.sas DDMMMYYYY HH:MM

#### Notes for Generating the Actual Table:

- n will be presented as an integer (with no decimal);
- Summary statistics will be presented with same precision as defined in post-text shells
- Internal template ITPar1, with the following changes: n will be presented in the column title with additional columns to be created.

For Table 12-2 through 12-5 the source tables will be 14.3.5.5

Program: /CAXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/adam intext pkparam.sas DDMMYYYY HH:MM

a - n = xx

<sup>\* -</sup> Single IV infusion of 0.25, 0.5 mg/kg xisomab 3G3 or placebo was administered on Day 1

Table 11-5 Summary of Kt/V Values (Safety Population)

| | Single pool Kt/V | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Treatments | | | | | | | | | | | | | |
| | Single IV Infusion of 0.25 mg/kg | | | | | | le IV Infu | sion of 0. | 5 mg/kg x | isomab | | Plac | cebo (Po | oled) | |
| Time | | X | cisomab | 3G3 | | | | 3G3 | | | | | | | |
| Point | R | t | UF | Wt | Kt/V | R | t | UF | Wt | Kt/V | R | t | UF | Wt | Kt/V |
| | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) |
| | [n=xx] | [n=xx] | [n=xx] | [n=xx] | [n=xx] | [n=xx] | [n=xx] | [n=xx] | [n=xx] | [n=xx] | [n=xx] | [n=xx] | [n=xx] | [n=xx] | [n=xx] |
| Day -7 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Day -5 | XX.X | XX.X | XX.X | XX.X <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Day -3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Day 1* | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Day 3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Day 5 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Day 12 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

a-n=xx

Values will be presented as arithmetic mean

R= post-dialysis BUN/pre-dialysis BUN))\*100

t = Time of HD

UF = Pre-dialysis Weight – Post-dialysis Weight

Wt = Post-dialysis weight of patient

 $Kt/V = ln(R - (0.008 \times t)) + (4 - (3.5 \times R)) \times \frac{UF}{Wt}$ 

Source: Tables 14.2.4.1.1 through 14.2.4.1.3

Program: /CAXXXXX/sas prg/stsas/intext/t ae.sas DDMMMYYYY HH:MM

#### Notes for Generating the Actual Table:

n will be presented as an integer (with no decimal);

- · Summary statistics will be presented with same precision as defined in post-text shells
- Internal template ITParl, with the following changes: n will be presented in the column title with more additional columns to be created.

Program: /CAXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMMYYYY HH:MM

Program: /CAXXXXX/sas prg/pksas/adam intext pkparam.sas DDMMYYYY HH:MM

<sup>\* -</sup> Single IV infusion of 0.25, 0.5 mg/kg xisomab 3G3 or placebo was administered on Day 1  $\,$
Table 11-7 Summary of Clotting in the Drip Chamber – Days -7 to 12 (Safety Population)

| | Clotting in the Drip Chamber Treatments | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | | T | reatm | ents | | | | | | | | | | | | | | |
| | S | Singl | e IV I | nfusio | n of 0.2 | 25 mg/ | kg xi | somab | 3G3 | | Sing | gle IV | Infus | ion of | 0.25 1 | ng/kg | xisor | nab 3 | G3 | | | | | Pla | icebo ( | Poole | ed) | | | |
| Time<br>Point | 2 H | ours | ategor<br>s after<br>Dialysi | Start | of | | | Catego<br>st-dial | • | | 2 | Hours | Catego<br>s after<br>Dialys | Start | of | | | atego<br>st-dia | | | 2 | Hour | Catego<br>s after<br>Dialys | r Start | of | | | Categ<br>ost-di | gory<br>alysis | |
| | | | [n=xx] | l | | | | [n=xx | ] | | | [n=xx] | | | | [n=xx] | | | | | [n=xy | x] | | | | [n=x | <b>x</b> ] | | | |
| | 1 | 2 | 3a | 3b | 4 | 1 | 2 | 3a | 3b | 4 | 1 | 2 | 3a | 3b | 4 | 1 | 2 | 3a | 3b | 4 | 1 | 2 | 3a | 3b | 4 | 1 | 2 | 3a | 3b | 4 |
| Day -7 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day -5 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day -3 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day 1* | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day 3 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day 5 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day 12 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day x | | | • | | | | | | | | | | | | | | | | | | | | | | | | | | | |

a-n=xx

Source: Table 14.2.6.1

Program: /CAXXXX/sas\_prg/stsas/intext/t\_ae.sas DDMMMYYYY HH:MM

### Notes for Generating the Actual Table:

- n will be presented as an integer (with no decimal);
- Summary statistics will be presented with same precision as defined in post-text shells
- Internal template ITParl, with the following changes: n will be presented in the column title with more additional columns to be created.

Program: /CAXXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMMYYYY HH:MM

Program: /CAXXXXX/sas prg/pksas/adam intext pkparam.sas DDMMMYYYY HH:MM

<sup>\* -</sup> Single IV infusion of 0.25, 0.5 mg/kg xisomab 3G3 or placebo was administered on Day 1 Values will be presented as arithmetic mean

Table 11-8 Summary of Clotting in the Dialysis Filter – Days -7 to 12 (Safety Population)

| | Clotting in Dialysis Filter Treatments | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Tr | eatme | nts | | | | | | |
| | S | Single | IV In | fusion | of | Sing | le IV | Infus | ion of | • | | Plac | ebo ( | Pooled | ) |
| | 0.2 | 5 mg | /kg xis | omab : | 3G3 | 0.25 | mg/k | g xiso | mab . | 3G3 | | | | | |
| Time<br>Point | | | Catego<br>ost-dia | • | | | | atego<br>st-dial | • | | | | Categ | • | |
| | | | [n=x | x] | | | | | | [n=x | x] | | | | |
| | 1 2 3a 3b 4 | | | | | 1 | 2 | 3a | 3 | 4 | 1 | 2 | 3a | 3b | 4 |
| | | | | | | | | | b | | | | | | |
| Day -7 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day -5 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day 1* | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day 3 | X X X X X X | | | X | X | X | X | X | X | X | X | X | X | X | |
| Day 5 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day 12 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Day x | | | | | | | | | | | | | | | |

a-n=xx

Source: Table 14.2.7.1

Program: /CAXXXXX/sas prg/stsas/intext/t ae.sas DDMMMYYYY HH:MM

### Notes for Generating the Actual Table:

- n will be presented as an integer (with no decimal);
- Summary statistics will be presented with same precision as defined in post-text shells
- Internal template ITPar1, with the following changes: n will be presented in the column title with more additional columns to be created.

Program: /CAXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYYY HH:MM

Program: /CAXXXXX/sas prg/pksas/adam intext pkparam.sas DDMMYYYY HH:MM

 $<sup>\</sup>ast$  - Single IV infusion of 0.25, 0.5 mg/kg xisomab 3G3 or placebo was administered on Day 1 Values will be presented as arithmetic mean

In-text Table 12-1 will be in the following format:

Table 12-1 Adverse Event Frequency by Treatment - Number of Subjects Reporting the Event (% of Subjects Dosed)

| | Dose Level of | xisomab 3G3 | Pooled | |
|---|---|---|---|---|
| Adverse Event* | 0.25 mg/kg | 0.5 mg/kg | Placebo | Overall |
| Number of Subjects With TEAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Number of Subjects Without TEAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| System Organ Class 1 | X (X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term 1 | X (X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term 2 | X (X%) | X (X%) | X (X%) | X (X%) |
| System Organ Class 2 | X (X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term 1 | X (X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term 2 | X (X%) | X (X%) | X (X%) | X (X%) |

\*Adverse events are classified according to MedDRA Version 21.1.

TEAEs = Treatment-emergent adverse events

If a subject has 2 or more clinical adverse events, the subject is counted only once within a category. The same subject may appear in different categories.

Source: Table 14.3.1.1

Program: /CAXXXXX/sas prg/stsas/intext/t\_ae.sas DDMMMYYYY HH:MM

### 11.2 Figures Shells

In-text Figures 11-1, 11-4 through 11-6, post-text Figures 14.2.1.2.1 through 14.2.1.2.3, 14.2.5.2.1 through 14.2.5.2.6 and Individual Listings in 16.2.6.1.1, 16.2.6.1.2, and 16.2.6.2.1 will be in the following format:

Figure 14.2.1.2.1

Arithmetic Mean (SD) Plasma Xisomab 3G3 Concentration Versus Time Profiles Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 (Linear Scale) (Pharmacokinetic Population)



Treatments B and C are shifted to the right for ease of reading Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

Figure 14.2.1.2.2

Arithmetic Mean Plasma Xisomab 3G3 Concentration Versus Time Profiles Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 (Linear Scale) (Pharmacokinetic Population)



Figure 14.2.1.2.3

Arithmetic Mean Plasma Xisomab 3G3 Concentration Versus Time Profiles Following a Single IV Infusion of 0.25 and 0.5 mg/kg Xisomab 3G3 (Semi-Log Scale) (Pharmacokinetic Population)



### Notes for Generating the Actual Mean Figure:

- Figures 11-1, 14.2.1.2.1 through 14.2.1.2.3
  - o y-axis: Plasma Xisomab 3G3 Concentration (ng/mL)
  - o X-axis: Hours From Start of Infusion
- Figures 11-4 and 11-5, 14.2.5.2.1 through 14.2.5.2.4
  - o y-axis: Arithmetic Mean aPTT (sec)
  - o X-axis: Hours From Start of Infusion
- Figures 11-6, 14.2.5.2.5 and 14.2.5.2.6
  - o y-axis: aPTT Mean Change from Baseline (sec)
  - o X-axis: Hours From Start of Infusion

Figure Legend: Use the Short Description as presented in Section 5.

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam meangraph.sas DDMMYYYY HH:MM

Figures 11-2, 11-3, 11-7, 14.2.2.2.1, 14.2.2.2.2, 14.2.3.2.1, 14.2.3.2.2, 14.2.5.2.7, and 14.2.5.2.8 will be listed as per the above formats with connecting the mean results between the pre- and post-dialysis results within the same day but without connecting the values between days.

oy-axis: <aPTT, Bun, potassium> (unit) o X-axis: Day

Figures in Appendices 16.2.6.1 and 16.2.6.2 will be in the following format:

Appendix 16.2.6.1.1 Individual Plasma Xisomab 3G3 Concentrations Versus Time Profiles Following a Single IV Infusion of <X> mg/kg Xisomab 3G3 (Linear and Semi-Log Scale) for Subject <#>



Program: /CAXXXXX/sas\_prg/pksas/adam\_indgraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/indgraph-all.sas DDMMMYYY HH:MM

### Notes for Generating the Actual Individual Figure:

- Appendix 16.2.6.1
  - o y-axis: Arithmetic Mean aPTT (sec)
  - o X-axis: Hours From Start of Infusion
- Appendix 16.2.6.2
  - o y-axis: Plasma Xisomab 3G3 Concentration (ng/mL)
  - o X-axis: Hours From Start of Infusion

Figure Legend: Use the Short Description as presented in Section 5.

Program: /CAXXXX/sas\_prg/pksas/indgraph-all.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_indgraph.sas DDMMYYYYY HH:MM

# 11.3 Section 14 Summary Tables Shells


Table 14.1.1 Subject Disposition Summary (Safety Population)

| | Dose Level of | Xisomab 3G3 | D 1 1 | |
|---|---|---|---|---|
| Disposition | 0.25 mg/kg | 0.5 mg/kg | - Pooled<br>Placebo | Overall |
| Dosed | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Completed | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Discontinued | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| <reason 1=""></reason> | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| <reason 2=""></reason> | X (XX%) | X (XX%) | X (XX%) | X (XX%) |

Program: /CAXXXXX/sas\_prg/stsas/tab PROGRAMNAME.sas DDMMYYYYY HH:MM

Table 14.1.2 Summary of Demographics (Safety Population)

| | | Dose Level of | | D 1 1 | |
|---|---|---|---|---|---|
| Trait | Category/<br>Statistics | 0.25 mg/kg | 0.5 mg/kg | Pooled<br>Placebo | Overall |
| Sex | Male<br>Female | | X ( XX%)<br>X ( XX%) | | , , |
| Race | Asian<br>Black or African<br>American<br>White | X ( XX%)<br>X ( XX%)<br>X ( XX%) | X ( XX%) | X (XX%) | X (XX%) |
| Ethnicity | Hispanic or Latino<br>Not Hispanic or Latino | | | X (XX%)<br>X (XX%) | , , |
| Age* (yrs) | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>XX.X<br>XX.XX<br>XX<br>XX.X<br>XX | X<br>XX.X<br>X.XX<br>XX<br>XX.X<br>XX | X<br>XX.X<br>X.XX<br>XX<br>XX<br>XX.X<br>XX | X<br>XX.X<br>X.XX<br>XX<br>XX<br>XX.X |
| Weight (kg) | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>XX.X<br>X.XX<br>XX<br>XX<br>XX.X | X<br>XX.X<br>X.XX<br>XX<br>XX.X<br>XX | X<br>XX.X<br>X.XX<br>XX<br>XX<br>XX.X<br>XX | X<br>XX.X<br>X.XX<br>XX<br>XX<br>XX.X |

Programmer Note: This is just a mock table shell. Please use the race categories listed in the CRF. Please also include Height (cm) and BMI (kg/m2).

Note: \*Age is calculated at the time of first dosing.

Program: /CAXXXXX/sas prg/stsas/tab PROGRAMNAME.sas DDMMMYYYY HH:MM

## Tables 14.2.1.1.1 through 14.2.1.1.3, 14.2.5.1.1 through 14.2.5.1.6 will be in the following format:

Table 14.2.1.1.1 Plasma Xisomab 3G3 Concentrations (ng/mL) Following a Single IV Infusion of 0.25 mg/kg Xisomab 3G3 (Pharmacokinetic Population)

| Subject | | | | Samp | ole Times | (hr) | | | |
|---|---|---|---|---|---|---|---|---|---|
| Number | Predose | XX | XX | XX | XX | XX | XX | XX | XX |
| X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX | XX | XX |

For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of  $<\!\!x\!>$  ng/mL are treated as 0 before the first quantifiable concentration and as missing elsewhere.

<sup>. =</sup> Value missing or not reportable.

#### Notes for Generating the Actual Table:

- Please use CPConc1 template
- Per study design needs, the following changes are made to this table relative to Celerion standard: columns <Treatment Sequence> and <Study Period> will be removed.
- Concentrations will be presented to the same precision as in the bio data.
- aPTT values will be presented to the same precision as in the clinical laboratory data.
- Summary statistics presentation with respect to the precision of the bio data or clinical laboratory data: n = integer; Mean and Median +1; SD and SEM +2, Minimum and Maximum +0, CV% to 1 decimal
- PK Time points are: predose (hour 0) and 0.167, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 96, 120, 144, and 192 hours postdose (additional time points might be added depending on the conduct of the study)
- For Tables 14.2.5.1.1 through 14.2.5.1.3, aPTT values will be reported during the course of the study from Days -7 through 12 with adding "Day" above the "Sampling Time".
- For Tables 14.2.5.1.3 and 14.2.5.1.6, there will be no summary statistics

Program: /CAXXXX/sas\_prg/pksas/pk-conc-tables.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/pk-conc-tables-sig.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam conc.sas DDMMYYYY HH:MM

Tables 14.2.1.1.4 and 14.2.1.1.5 will be in the following format:

Table 14.2.1.1.4 Plasma Xisomab 3G3 Pharmacokinetic Parameters Following a Single IV Infusion of 0.25 mg/kg Xisomab 3G3 (Pharmacokinetic Population)

| | | | P | Parameters | | |
|---|---|---|---|---|---|---|
| Subject | param1 | param2 | param3 | param4 | param5 | param6 |
| | (units) | | | | | |
| | XXX | | | | XX.X | |
| X | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| X | X.XX | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XXX | | | | XX.X | |
| n | XX | | XX | | XX | |
| Mean | XXX.X | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| Median | XX.XX | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| Maximum | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| Geom Mean | XXX.X | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| Geom CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

. = Value missing or not reportable.

#### Notes for Generating the Actual Table:

- Please use CPPar1 template
- Per study design needs, the following changes are made to this table relative to Celerion standard: columns <Treatment Sequence> and <Study Period> will be removed.
- PK Parameters will be presented in the following order and with following units: AUCO-t <ng\*hr/mL>, AUCO-inf <ng\*hr/mL>, AUC%extrap <%>, Cmax <ng/mL>, Tmax <hr>, Kel <1/hr>, T1/2 <hr>, CL <L/hr>, Vss <L>
- n will be presented as an integer (with no decimal);
- Exposure parameters (i.e. AUCs, Cmax, Vss, CL) will be presented with, at maximum, the precision of the bio data, and, at minimum, 3 significant figures (to be determined by the PKist once bio data are received).
  - o Summary statistics will be presented with respect to the precision of the bio data: Mean, Median, and Geom Mean = +1; SD and SEM = +2, Minimum and Maximum = +0.
- Time parameters (i.e. Tmax, t1/2) will be presented with 2 decimals.
  - o Summary statistics will be presented with respect to the number of decimals: Mean, Median, and Geom Mean = +1; SD and SEM = +2, Minimum and Maximum = +0.
- Values for rate constants (i.e. Kel) will be presented with 3 significant figures.
  - o Summary statistics for Kel will be presented as: Mean, Median, and Geom Mean = +1; SD and SEM = +2, Minimum and Maximum = +0.
- CV% and Geom CV% for all parameters will be presented with 1 decimal

Program: /CAXXXX/sas\_prg/pksas/pk-tables.sas DDMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam pkparam.sas DDMMYYYY HH:MM

## Table 14.2.1.1.6 will be in the following format:

Table 14.2.1.1.6 Intervals (Hours) Used for Determination of Plasma Xisomab 3G3 Kel Values (Pharmacokinetic Population)

| Subject<br>Number | Treatment | Interval | R2 | n |
|-------------------|------------|-------------|-------|---|
| <br>X | 0.25 mg/kg | xx.x - xx.x | X.XXX | X |
| X | 0.5 mg/kg | XX.X - XX.X | X.XXX | X |
| X | X | XX.X - XX.X | X.XXX | X |
| X | X | XX.X - XX.X | X.XXX | X |
| X | X | XX.X - XX.X | X.XXX | X |
| X | X | XX.X - XX.X | X.XXX | X |

0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

R2 = Coefficient of determination

n = Number of points used in Kel calculation

. = Kel value not reportable.

#### Notes for Generating the Actual Table:

- Please use CPKel1 template
- Per study design, the "Treatment Sequence" column will be replaced with 'Treatment" and the data will be presented vertically instead of horizontally.
- Interval start and stop times will be presented to 1 decimal or 3 significant figures minimum
- R2 will be presented to 3 decimals
- n will be presented as an integer

Program: /CAXXXXX/sas\_prg/pksas/kel-tables-xover.sas DDMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam kel.sas DDMMYYYY HH:MM

Tables 14.2.2.1.1 through 14.2.2.1.3, 14.2.3.1.1 through 14.2.3.1.3 will have the following format:

Table 14.2.3.1.1 Individual and Mean Difference Between Pre- and Post-dialysis Potassium Values (unit) - Days -7 to 12 - 0.25 mg/kg Xisomab 3G3 on Day 1 (Safety Population)

| | | | 0.25 m | g/kg | | | 0.5 mg/kg | | | | Placebo | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Day | Pre-<br>dialysis<br>(units) | Post-<br>dialysis<br>(units) | Differ<br>(un | ence | Pre-<br>dialysis<br>(units) | Post-<br>dialysis<br>(units) | Di | ifference<br>(units) | Pre-<br>dialysis<br>(units) | Post-<br>dialysis<br>(units) | Difference (units) |
| X | _ | 7 XX | XX X. | | | | XX XX | . X | X.XXX | XXX | XX.X | X.XXX |
| X | - | 7 XX. | XX.X X.XX XXX | | | XXX XXX | XX XX | . X | X.XXX | XXX | XX.X | X.XXX |
| X | - | 7 XX. | Х Х. | X.XX XXX | | XXX XXX | XX XX | . X | X.XXX | XXX | XX.X | X.XXX |
| X | - | 7 X.X | XX X. | XX | XXX | XXX XXX | XX XX | . X | X.XXX | XXX | XX.X | X.XXX |
| X | - | 7 XX | XX X. | XX | XXX | XXX XXX | XX XX | . X | X.XXX | XXX | XX.X | X.XXX |
| n | | Σ | X | XX | XX | X | | XX | XX | XX | XX | XX |
| Mean | | XXX. | X X.X | XXX | XXX.X | XXX. | XX. | XX | X.XXXX | XXX.X | XX.XX | X.XXXX |
| SD | | XX.X | XX XX. | XX | XX.XX | XX.XX | XX. | XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | XX. | X XX | Χ.Χ | XX.X | XX.X | XX XX | . X | XX.X | XX.X | XX.X | XX.X |
| SEM | | XX.X | XX XX. | XX | XX.XX | XX.XX | XX. | XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | | XX. | Х Х. | XX | XXX | XXX XXX | XX X | . X | X.XXX | XXX | XX.X | X.XXX |
| Median | | XX.X | XX X.X | XXX | XXX.X | XXX. | XX. | XX | X.XXXX | XXX.X | XX.XX | X.XXXX |
| Maximum | | XX | XX X. | XX | XXX | XXX | XX XX | . X | X.XXX | XXX | XX.X | X.XXX |

0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

Placebo = pooled placebo

Difference = Pre-dialysis - Post-dialysis

Single IV infusion of 0.25, 0.5 mg/kg xisomab 3G3 or placebo was administered on Day 1

#### Programmer Notes:

For the BUN Tables 14.2.2.1.1 through 14.2.2.1.3 values will be reported at pre- and post-dialysis on Days -7, -5, -3, 1, 3, 5, 6, and 12. The screening values to be reported if not presented in other tables.

For the BUN Tables 14.2.2.1.1 through 14.2.2.1.3, additional column of "URR" will be reported at the right of the "Difference" column (as per Table 11-3 shell), with the following footnotes:

- Difference = Pre-dialysis Post-dialysis
- ullet Single IV infusion of 0.25, 0.5 mg/kg xisomab 3G3 or placebo was administered on Day 1
- URR = (1-(post-dialysis BUN/ pre-dialysis BUN))\*100

Program: /CAXXXX/sas\_prg/pksas/xxxxxxxx.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/xxxxxxxxx.sas DDMMYYYY HH:MM

Tables 14.2.5.1.7 through 14.2.5.1.9, 14.2.4.1.1 through 14.2.4.1.3 will have the following format:

Table 14.2.5.1.7 Individual and Mean Difference Between Pre- and Post-dialysis aPTT Values (unit) - Days -7 to 12 - 0.25 mg/kg Xisomab 3G3 on Day 1 (Safety Population)

| | | | 0.25 mg/kg | | 0 | .5 mg/kg | | | Placebo | · |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Day | Pre-<br>dialysis<br>(units) | Post-<br>dialysis<br>(units) | Fold<br>Change<br>(units) | Pre-<br>dialysis<br>(units) | Post-<br>dialysis<br>(units) | Fold<br>Change<br>(units) | Pre-<br>dialysis<br>(units) | Post-<br>dialysis<br>(units) | Fold<br>Change<br>(units) |
| X | -7 | XXX | X.XX | XXX | XXX | XX.X | X.XXX | XXX | XX.X | X.XXX |
| X | -7 | XX.X | X.XX | XXX | XXX | XX.X | X.XXX | XXX | XX.X | X.XXX |
| X | -7 | XX.X | X.XX | XXX | XXX | XX.X | X.XXX | XXX | XX.X | X.XXX |
| X | -7 | X.XX | X.XX | XXX | XXX | XX.X | X.XXX | XXX | XX.X | X.XXX |
| X | -7 | XXX | X.XX | XXX | XXX | XX.X | X.XXX | XXX | XX.X | X.XXX |
| n | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | | XXX.X | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX | XXX.X | XX.XX | X.XXXX |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | | XX.X | X.XX | XXX | XXX | XX.X | X.XXX | XXX | XX.X | X.XXX |
| Median | | XX.XX | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX | XXX.X | XX.XX | X.XXXX |
| Maximum | | XXX | X.XX | XXX | XXX | XX.X | X.XXX | XXX | XX.X | X.XXX |

0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3

 $0.5~\mathrm{mg/kg}\colon \mathrm{Single}\ \mathrm{IV}\ \mathrm{Infusion}$  of  $0.5~\mathrm{mg/kg}\ \mathrm{xisomab}\ 3\mathrm{G3}$ 

Placebo = pooled placebo

Fold Change = Post-dialysis / Pre-dialysis

Single IV infusion of 0.25, 0.5 mg/kg xisomab 3G3 or placebo was administered on Day 1

#### Programmer Notes:

Values will be reported at pre- and post-dialysis on Days -7, -5, -3, 1, 3, 5, 6, and 12. The screening values to be reported if not presented in other tables.

For Tables 14.2.4.1.1 through 14.2.4.1.3, Kt/V will be reported on Days -7, -5, -3, 1, 3, 5, and 12. Column titles will be the same as per Table 11-5 shell (ie., R, t, UF, Wt, and Kt/V) with the following footnotes:

- Single IV infusion of 0.25, 0.5 mg/kg xisomab 3G3 or placebo was administered on Day 1
- R = post-dialysis BUN/pre-dialysis BUN))\*100
- t = Time of HD
- UF = Pre-dialysis Weight Post-dialysis Weight
- Wt = Post-dialysis weight of patient
- Kt/V =  $ln(R (0.008 \times t)) + (4 (3.5 \times R)) \times \frac{UF}{Wt}$

For the bleeding time table in Section 14.3, values will be reported post-dialysis on Days screening (if available), -7, -5, -3, 1, 3, 5, 8, 10 and 12. There will be only one column underneath each dose as per Table 11-4 shell with the following footnote:

• Single IV infusion of 0.25, 0.5 mg/kg xisomab 3G3 or placebo was administered on Day 1

Program: /CAXXXX/sas\_prg/pksas/xxxxxxxx.sas DDMMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/xxxxxxxxx.sas DDMMMYYYY HH:MM

Tables 14.2.6.1 will be in the following format:


Table 14.2.6.1 Summary of Clotting in the Drip Chamber - Days -7 to 12 (Safety Population)

| | | 0.2 | 5 mg | /kg X | isomab | 3G3 | 0. | 5 mg | r/kg X | isomal | o 3G3 | Po | oole | d Plac | cebo | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Catego | ory* | | | Cat | egory | * | | | Cat | egor | У* | |
| Day | Time Point | 1 | 1 2 3a 3b 4 | | | 1 | 2 | 3a | 3b | 4 | 1 | 2 | 3a | 3b | 4 | |
| <br>Day -7 | 2 hr after HD | Х | X | Х | Х | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | Post HD | X | Х | Х | Х | Х | Х | Х | Х | Χ | Χ | Χ | Х | Х | Х | Х |
| Day X | 2 hr after HD | Х | Х | Х | Χ | Х | Х | Х | Х | Χ | X | Х | Х | Х | Χ | Х |
| | Post HD | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х |

<include all days and timepoints>

Note: \*Category:1=No detectable clotting, 2=Presence of fibrinous ring or minimum clot affecting less than 5% of chamber space, 3a=Clot formation (affecting more than 5% of but less than 30% of chamber space) but dialysis still possible, 3b=Clot formation (affecting more than 30% of chamber space) but dialysis still possible,

4=Complete occlusion of chamber

HD: hemodialysis

Program: /AAXXXXX/ECR/sas prg/stsas/tab PROGRAMNAME.sas DDMMMYYYY HH:MM

Tables 14.2.7.1 will be in the following format:

Table 14.2.7.1 Summary of Clotting in the Dialysis Filter - Days -7 to 12 (Safety Population)

| | | 0.2 | 5 mg/ | kg X | isomab | 3G3 | 0.5 mg/kg Xisomab 3G3 | | | | | Po | oole | d Plac | cebo | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | ( | Catego | ory* | | | Cat | egory | * | | | Cat | egory | <u>/</u> * | |
| | Day | 1 | 2 | 3a | 3b | 4 | 1 | 2 | 3a | 3b | 4 | 1 | 2 | 3a | 3b | 4 |
| - | Day -7 | X | X | Х | X | X | X | Х | Х | X | Х | X | Χ | Х | Х | X |
| | Day X | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |

<include all days>

Note: \*Category:1= No clotting, clean filter, 2= Few blood streaks (affecting less than 5% of the fibers seen at the surface of dialyzer),
3a= More blood streaks (affecting more than 5% but less than 30 % of the fibers seen at the surface of the dialyzer),
3b= More blood streaks (affecting more than 30% of the fibers seen at the surface if the dialyzer),
4=Complete occlusion

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMYYYYY HH:MM


Table 14.3.1.1 Treatment-Emergent Adverse Event Frequency by Treatment - Number of Subjects Reporting the Event (% of Subjects Dosed) (Safety Population)

| | | f Xisomab 3G3 | D 1 1 | |
|---|---|---|---|---|
| Adverse Event* | | 0.5 mcg/kg | Pooled<br>Placebo | Overall |
| Number of Subjects Dosed<br>Number of Subjects With TEAEs^<br>Number of Subjects Without TEAEs^ | , , | XX (XXX%)<br>X ( XX%)<br>XX (XXX%) | X ( XX%) | , , |
| Nervous system disorders Dizziness Headache Presyncope Respiratory, thoracic and mediastinal disorders Dry throat Oropharyngeal pain Sinus congestion Sneezing | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| General disorders and administration site conditions Fatigue Thirst | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |

Note: \*Adverse events are classified according to MedDRA Version 21.1. ^ = Treatment-emergent adverse events

If a subject has 2 or more clinical adverse events, the subject is counted only once within a category. The same subject may appear in different categories.

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMYYYYY HH:MM

Table 14.3.1.2 Treatment-Emergent Adverse Event Frequency by Treatment - Number of Adverse Events (% of Total Adverse Events) (Safety Population)

| | Dose Level c | | | |
|---|---|---|---|---|
| Adverse Event* | | 0.5 mg/kg | | Overall |
| Number of TEAEs | X (100%) | X (100%) | X ( XX%) | X ( XX%) |
| Nervous system disorders | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Dizziness | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Headache | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Presyncope | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Respiratory, thoracic and mediastinal disorders | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Dry throat | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Oropharyngeal pain | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Sinus congestion | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Sneezing | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| General disorders and administration site | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| conditions | | | | |
| Fatique | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Thirst | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |

Note: \*Adverse events are classified according to MedDRA Version 21.1. ^ = Treatment-emergent adverse events

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Table 14.3.1.3 Treatment-Emergent Adverse Event Frequency by Treatment, Severity, and Relationship to Study Drug - Number of Adverse Events (Safety Population)

| | | | Severity | | | | | Relationship to Study Drug | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event* | Dose<br>Level/<br>Placebo | Number of<br>Subjects<br>With TEAEs | Number<br>of<br>TEAEs | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Unrelated | Unlikely | Possibly | Probably | Likely |
| Dizziness | X | X | Х | X | X | Х | Х | X | X | X | Х | X |
| | X | X | X | X | X | X | X | X | X | X | X | X |
| Dry eye | X | X | X | X | X | X | X | X | X | X | X | X |
| Dry mouth | X | X | X | X | X | X | X | X | X | X | X | X |
| Dry throat | X | X | X | X | X | X | X | X | X | X | X | X |
| Ear pain | X | X | X | X | X | X | X | X | X | X | X | X |
| | X | X | X | X | X | X | X | X | X | X | X | X |
| Fatigue | X | X | X | X | X | X | X | X | X | X | X | X |
| Headache | X | X | X | X | X | X | X | X | X | X | X | X |
| Dizziness | X | X | X | X | X | X | X | X | X | X | X | X |
| | X | X | X | X | X | X | X | X | X | X | X | X |
| Hyperhidrosis | X | X | X | X | X | X | X | X | X | X | X | X |
| Laceration | X | X | X | X | X | X | X | X | X | X | X | X |
| Limb crushing injury | X | X | X | X | X | X | X | X | X | X | X | X |
| Muscle twitching | Χ | X | X | X | X | X | X | X | X | X | X | X |
| 0.25 m | ng/kg | X | X | X | X | Х | X | X | X | X | X | X |
| 0.5 m | | X | X | X | X | X | X | X | X | X | X | X |
| | acebo | XX | XX | X | X | X | X | X | X | X | X | X |
| Ove | erall | XX | XX | X | X | X | X | X | X | X | X | X |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3

0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

Placebo = pooled placebo

\*Adverse events are classified according to MedDRA Version 21.1. TEAE = Treatment-emergent adverse events

If a subject experience the same adverse event (AE) at more than one level of severity during a treatment, each AE is counted separately. If a subject experience the same AE at more than one level of drug relationship during a treatment, each AE is counted separately.

Severity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially life-threatening

Program: /CAXXXXX/sas prg/stsas/tab PROGRAMNAME.sas DDMMMYYYY HH:MM

Tables 14.3.4.1 to 14.3.4.3 will have the following format:


Table 14.3.4.1 Out-of-Range Values and Clinically Significant Results - Serum Chemistry (Safety Population)

| | | | | | | | | Parameter1 | Parameter2 | Parameter3 | Parameter4 | Parameter5 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose Level/ | Subject | : Age#/ | Study | | | | | <range></range> | <range></range> | <range></range> | <range></range> | <range></range> |
| Placebo | Number | Sex | Period | Day | Hour | Date | Time | (Unit) | (Unit) | (Unit) | (Unit) | (Unit) |
| XXX <units></units> | X | XX/X | Screen | | • | DDMMYYYYY | HH:MM:SS | XX H + | | | | XX L |
| | | | 1 | -X | -XX.XX | DDMMYYYY | HH:MM:SS | XX L | XX L | XX H | XX L | |
| | | | Recheck | | | DDMMYYYYY | HH:MM:SS | | | | XX | |

Programmer Notes: Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early termination

chronologically with other scheduled assessments.

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3

0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3  $\,$ 

Placebo = pooled placebo

#Age is calculated at the time of first dosing. F = Female; M = Male

H = Above reference range, L = Below reference range

PI Interpretation: + = Clinically significant

Program: /CAXXXX/sas prg/stsas/tab PROGRAMNAME.sas DDMMYYYY HH:MM

## Tables 14.3.5.1, 14.3.5.3 and 14.3.5.5 will be in the following format:


Table 14.3.5.1 Clinical Laboratory Summary and Change from Baseline - Serum Chemistry (Safety Population)

| | | | | | Change from Baseline* | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Laboratory Test (unit) | Reference<br>Range | Time Point | Statistic | 0.25<br>mg/kg | 0.5<br>mg/kg | Placebo | 0.25<br>mg/kg | 0.5<br>mg/kg | Placebo |
| XXXXXXXXX (unit) | X.X-XX.X# | Screen | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>X.XX<br>X.XXX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XX<br>X.XX<br>X.X | | | |
| | | Baseline* | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>X.XX<br>X.XX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XX<br>X.X | | | |
| | | Day X, Hour X.XX | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>X.XX<br>X.XX<br>X.X<br>X.X | XX<br>X.XX<br>X.XX<br>X.X<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XX<br>X.XX<br>X.X<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XX<br>X.XX<br>X.X<br>X.X |

#### <include all timepoints>

Programmer Note: Table 14.3.5.5 will not include timepoints that are summarized in PD endpoint tables in 14.2.

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3

0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

Placebo = pooled placebo

- # = Lowest of the lower ranges and highest of the higher ranges are used. Refer to Appendix 16.1.10.1 for the breakdown.
- \* Baseline is defined as the result closest and prior to dose on Day 1.

Programmer note: for PT, INR and PT/INR, the pre-dialysis value will be the baseline value for that day and the "change from baseline" will be the fold change from baseline "ie. Post-dialysis / Pre-dialysis.

Program: /AAXXXXX/ECR/sas prg/stsas/tab PROGRAMNAME.sas DDMMMYYYY HH:MM

## Tables 14.3.5.2, 14.3.5.4 and 14.3.5.6 will be in the following format:


Table 14.3.5.2 Clinical Laboratory Shift From Baseline - Serum Chemistry (Safety Population)

| Taboratory Test | Dose<br>Level/ | | Baseline* L | | | Baseline* N | | | Baseline* H | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| (unit) | Placebo | Time Point | L | N | Н | L | N | Н | L | N | Н |
| XXXXXXX (unit) | XXX <units></units> | Day X, Hour X.XX | X | XX | X | X | XX | X | X | XX | X |

Programmer Note: Table 14.3.5.6 will not include timepoints that are summarized in PD endpoint tables in 14.2.

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3

0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

Placebo = pooled placebo

N = Within Normal Range, L = Below Normal Range, H = Above Normal Range

# = Lowest of the lower ranges and highest of the higher ranges are used. Refer to Appendix 16.1.10.1 for the breakdown.

\* Baseline is defined as the result closest and prior to dose on Day 1.

Program: /AAXXXX/ECR/sas prg/stsas/tab PROGRAMNAME.sas DDMMYYYY HH:MM

Table 14.3.5.7 Vital Sign Summary and Change from Baseline (Safety Population)

| | | | | | | Chang | Change from Baseline* | |
|---|---|---|---|---|---|---|---|---|
| Vital Sign(unit) | Time Point | Statistic | 0.25<br>mg/kg | 0.5<br>mg/kg | Placebo | 0.25<br>mg/kg | 0.5<br>mg/kg | Placebo |
| XXXXXXXXX (unit) | Screen | n | XX | XX | XX | | | |
| | | Mean | X.XX | X.XX | X.XX | | | |
| | | SD | X.XXX | X.XXX | X.XXX | | | |
| | | Minimum | X.XX | X.XX | X.XX | | | |
| | | Median | X.X | X.X | X.X | | | |
| | | Maximum | XX.X | XX.X | XX.X | | | |
| | <also -3="" -5="" -7,="" and="" days="" include=""></also> | | | | | | | |
| | Baseline* | n | XX | XX | XX | | | |
| | | Mean | X.XX | X.XX | X.XX | | | |
| | | SD | X.XXX | X.XXX | X.XXX | | | |
| | | Minimum | X.XX | X.XX | X.XX | | | |
| | | Median | X.X | X.X | X.X | | | |
| | | Maximum | XX.X | XX.X | XX.X | | | |
| | Day X, Hour X.XX | n | XX | XX | XX | XX | XX | XX |
| | , | Mean | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | SD | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| | | Minimum | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Median | | X.X | X.X | X.X | X.X | X.X |
| | | Maximum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

#### <include all postdose timepoints>

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo

\* Baseline is defined as the result closest and prior to the dose on Day 1.

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMYYYY HH:MM

Table 14.3.5.8 12-Lead Electrocardiogram Summary and Change from Baseline (Safety Population)

| | | | | | | Chang | Change from Baseline* | |
|---|---|---|---|---|---|---|---|---|
| Measurement (unit) | Time Point | Statistic | | 0.5<br>mg/kg | Placebo | 0.25<br>mg/kg | | Placebo |
| XXXXXXXXX (unit) | Screen | n | XX | XX | XX | | | |
| , , | | Mean | X.XX | X.XX | X.XX | | | |
| | | SD | X.XXX | X.XXX | X.XXX | | | |
| | | Minimum | X.XX | X.XX | X.XX | | | |
| | | Median | X.X | | X.X | | | |
| | | Maximum | XX.X | XX.X | XX.X | | | |
| | Baseline* | n | XX | XX | XX | | | |
| | | Mean | X.XX | X.XX | X.XX | | | |
| | | SD | X.XXX | X.XXX | X.XXX | | | |
| | | Minimum | X.XX | X.XX | X.XX | | | |
| | | Median | X.X | X.X | X.X | | | |
| | | Maximum | XX.X | XX.X | XX.X | | | |
| | Day X, Hour X.XX | n | XX | XX | XX | XX | XX | XX |
| | , | Mean | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | SD | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| | | Minimum | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Median | X.X | | X.X | X.X | X.X | X.X |
| | | Maximum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

#### <include all postdose timepoints>

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

Placebo = pooled placebo

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMYYYY HH:MM

Tables 14.2.12 will be in the following format:

 $<sup>^{\</sup>star}$  Baseline is defined as the result closest and prior to the dose on Day 1.


Table 14.5.5.9 Frequency of Immunogenicity - ADA Titer (Safety Population)

| | 0.25 mg/kg 1 | Kisomab 3G3 | 0.5 mg/kg | Xisomab 3G3 | Pooled Placebo | |
|---|---|---|---|---|---|---|
| Day | Positive | Negative | Positive | Negative | Positive | Negative |
| Day 1 | X (%) | X (%) | X (%) | X (%) | X (%) | X (%) |
| Day 12 | X (%) | X (%) | X (%) | X (%) | X (%) | X (%) |

Note: % is percentage of total subject dosed in each treatment.

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMYYYYY HH:MM

### 12. LISTING SHELLS

The following listing shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the listings that will be presented and included in the final CSR. These listings will be generated off of the Celerion SDTM Tabulation Model 1.4 mapped in accordance with SDTM Implementation Guide 3.2. All listings will be presented in Courier New size font 9.

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

| Laboratory Group | Test Name | Sex | Age Category | Reference<br>Range | Unit |
|---|---|---|---|---|---|
| Serum Chemistry | Test Name | XXXXXX | XX | XX - XX | units |
| _ | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| Hematology | Test Name | XXXXXX | XX | xx - xx | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |

<similar for remaining Laboratory Groups and Test Names>

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Appendix 16.2.1 Study Completion/Early Termination (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | | Date | Date of<br>Last Contact | Reason for Discontinuation | Comments |
|---|---|---|---|---|---|---|
| XXX <units></units> | Х | Yes | DDMMYYYYY | DDMMYYYY | | |
| | X | Yes | DDMMYYYYY | DDMMYYYYY | | |
| | X | Yes | DDMMYYYYY | DDMMYYYYY | | |
| | X | Yes | DDMMYYYYY | DDMMYYYYY | | |
| | X | No | DDMMYYYYY | DDMMYYYYY | XXXXXXXXXXXXX | XXXXXXX |
| | X | Yes | DDMMYYYYY | DDMMYYYYY | | |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo

Program: /AAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Appendix 16.2.4.1 Demographics (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | Date of<br>Birth | Age*<br>(yrs) | Sex | Race | Ethnicity | Height<br>(cm) | Weight<br>(kg) | Body Mass<br>Index<br>(kg/m²) | Informed<br>Consent<br>Date |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX <units></units> | X | MMYYYY | XX | AAAAAA | AAAAAAA | AAAAAAAA | XXX | XX.XX | XX.XX | DDMMYYYY |
| | X | MMMYYYY | XX | AAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DDMMYYYYY |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo

\*Age is calculated from the date of first dosing.

Program: /AAXXXXX/sas prg/stsas/lis PROGRAMNAME.sas DDMMMYYYY HH:MM

#### Appendix 16.2.4.2 Physical Examination (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | | Day | Time | Date | Body System | Result | Abnormality | Clinical<br>Significance |
|---|---|---|---|---|---|---|---|---|---|
| XXX <units></units> | Х | Screen | | | DDMMYYYY | 1. General Appearance | Abnormal | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | NCS |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.4.3 Medical and Surgical Histories (Safety Population)

| Dose Level/ | Subject | | | Date of Diagno | | |
|---|---|---|---|---|---|---|
| Placebo | | | Description | Start | End | Ongoing? |
| XXX <units></units> | X | Х | XXXXXX XXXXXX XXXXXXX | DDMMYYYYY | | Yes |
| | | X | XXXXXXXX | DDMMYYYYY | DDMMYYYYY | No |
| | | X | XXXXXXXX XXXXXX XXXXXX | DDMMYYYYY | DDMMMYYYY | No |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.4.4 Alcohol Screen (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | Visit<br>Date | Type of Sample | Actual<br>Time | Result |
|---|---|---|---|---|---|
| XXX <units></units> | X | DDMMYYYYY | Urine | HH:MM | Negative |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.4.5 Drug Screen (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | Visit<br>Date | Type of Sample | Actual<br>Time | Result | If Positive, | list all | that were positive: |
|---|---|---|---|---|---|---|---|---|
| XXX <units></units> | × | DDMMMYYYY | Urine | <br>HH•MM | Negative | | | |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.5.1 Subject Eligibility (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | | Date | Did subject meet all eligibility criteria? | Criterion Not Met* | Specify |
|---|---|---|---|---|---|---|
| XXX <units></units> | X<br>X | Screen<br>Screen | DDMMYYYY<br>DDMMYYYY | Yes<br>Yes | | |
| | X | Screen | DDMMYYYY | No | EXCLUSION X | XXXXXXXXXXXXXXX XXXX |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.5.2 Subject Eligibility at Check-In (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | - | Date | Does subject continue to meet criteria since Screening? | If No, specify |
|---|---|---|---|---|---|
| XXX <units></units> | X | Check-In | DDMMYYYY | Yes | |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


#### Appendix 16.2.5.3 Test Compound Administration Times (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | Period | Day | Time | Dose<br>Date | Start<br>Administered? | End<br>Time | Time | Route | Form | Frequency |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX <units></units> | X | XXXX | XX | XX | DDMMYYYY | Yes | HH:MM:SS | HH:MM:SS | IV Infusion | Injection | Once |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.5.4 Blood Draw Times for Free XISOMAB 3G3 PK (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | Day | Hour | Date | Actual<br>Time | Comments |
|---|---|---|---|---|---|---|
| XXX <units></units> | X | Х | -X.XX<br>XX.XX<br>XX.XX | DDMMYYYY<br>DDMMYYYY<br>DDMMYYYY | XX:XX<br>XX:XX<br>XX:XX | XXXXXXXXXX |
| | | | XX.XX<br>XX.XX<br>XX.XX | DDMMYYYY<br>DDMMYYYY<br>DDMMYYYY | XX:XX<br>XX:XX<br>XX:XX | XXXXXXXXX |
| | | | XX.XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | DDMMYYYY DDMMYYYY DDMMYYYY DDMMYYYY DDMMYYYY DDMMYYYY | XX:XX<br>XX:XX<br>XX:XX<br>XX:XX<br>XX:XX<br>XX:XX | XXXXXXXXXX |
| | | Х | XX.XX | DDMMMYYYY | XX:XX | |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.5.5 Blood Draw Times for Free XISOMAB 3G3 PD (aPTT) (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | Day | Hour | Date | Actual<br>Time | Comments |
|---|---|---|---|---|---|---|
| XXX <units></units> | Х | X | -X.XX<br>XX.XX<br>XX.XX | DDMMMYYYY<br>DDMMMYYYY | XX:XX<br>XX:XX<br>XX:XX | XXXXXXXXXX |
| | | | XX.XX<br>XX.XX<br>XX.XX | DDMMYYYY<br>DDMMYYYYY<br>DDMMYYYYY | XX:XX<br>XX:XX<br>XX:XX | XXXXXXXXX |
| | | | XX.XX<br>XX.XX<br>XX.XX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | XX:XX<br>XX:XX<br>XX:XX | XXXXXXXXXX |
| | | X | XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | XX:XX<br>XX:XX<br>XX:XX<br>XX:XX | |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.5.6 Blood Draw Times for Immunogenicity (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | Day | Hour | Date | Actual<br>Time | Comments |
|---|---|---|---|---|---|---|
| XXX <units></units> | X | _ | Predose<br>Follow-up | | HH:MM<br>HH:MM | XXXXXXXXXX |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.5.7 Blood Draw Times for Dialysate Analysis for Kt/V and URR (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | Day | Hour | Date | Actual<br>Time | Comments |
|---|---|---|---|---|---|---|
| XXX <units></units> | X | <del>-</del> 7 | 3 hours | DDMMYYYY | HH:MM | XXXXXXXXXX |
| | | <b>-</b> 5 | 3 hours | DDMMYYYYY | HH:MM | |
| | | 1 | 3 hours | DDMMYYYY | HH:MM | |
| | | 3 | 3 hours | DDMMYYYY | HH:MM | |
| | | 12 | 3 hours | DDMMYYYYY | HH:MM | |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.5.8.1 Dialyzer Assessment (I of V) (Safety Population)

| Dose Level/ | Subject | | | Hemodialys | | Interrupted | | |
|---|---|---|---|---|---|---|---|---|
| Placebo | _ | | Day | Start End | Total* | _ | Reason for Interruption | Specify |
| XXX <units></units> | Х | XXXX | Х | HH:MM HH:MM | HH:MM | Yes | | = |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo \*Total = End time - Start time


Appendix 16.2.5.8.2 Dialyzer Assessment (II of V) (Safety Population)

| | | | | | | | | Blood | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Atrial | Pressure | Venus P | ressure | Flow | Time t | o Hemost | asis | |
| Dose Level/ | Subject | | | | | | | Rate | | | | Dialysis Filter |
| Placebo | Number | Day | Hour | Time | mmHg | Time | mmHg | mL/min | Time | Length | (min) | Collected*? |
| XXX <units></units> | Y | Y | Y | HH • MM | XX | HH • MM | XX | XX | HH • MM | XX | | Yes |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

Placebo = pooled placebo

<sup>\*</sup> Was the dialysis fi lter collected, sealed and stored < -20 C until shipment?


Appendix 16.2.5.8.3 Dialyzer Assessment (III of V) - Number and Volume of Saline Flushes (Safety Population)

| Dose Level/<br>Placebo | Subject<br>Number | Day | Hour | Saline<br>Flush<br>Number | of | Volume<br>(mL) | Total Volume<br>of Flushes (mL) | Total Number<br>of Flushes |
|---|---|---|---|---|---|---|---|---|
| XXX <units></units> | X | X | X | 1<br>2<br>3<br>4<br>5 | HH:MM<br>HH:MM<br>HH:MM<br>HH:MM<br>HH:MM | XX<br>XX<br>XX<br>XX<br>XX<br>XX | XXX | XX |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.5.8.4 Dialyzer Assessment (IV of V) - Clotting in the Drip Chamber (Safety Population)

| | | | | 2 Hours | afte | er St | tart | of D | ialys | is | | I | End o | of Di | alys: | is |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose Level/ | Subject | | | | | Ca | atego | ry* | | | | | Cá | atego | ry* | |
| | Number | Day | Hour | Time | 1 | 2 | 3a | 3b | 4 | | Time | 1 | 2 | 3a | 3b | 4 |
| XXX <units></units> | × | × | х | HH • MM | × | X | | | | <b></b> - | <br>нн • мм | | <u>-</u> - | | | <b>-</b> - |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

Placebo = pooled placebo

\*Category:1=No detectable clotting, 2=Presence of fibrinous ring or minimum clot affecting less than 5% of chamber space, 3a=Clot formation (affecting more than 5% of but less than 30% of chamber space) but dialysis still possible, 3b=Clot formation (affecting more than 30% of chamber space) but dialysis still possible, 4=Complete occlusion of chamber


Appendix 16.2.5.8.5 Dialyzer Assessment (V of V) - Clotting in Dialysis Filter (Safety Population)

## End of Dialysis (or premature interruption)

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

Placebo = pooled placebo

\*Category:1= No clotting, clean filter, 2= Few blood streaks (affecting less than 5% of the fibers seen at the surface of dialyzer),
3a= More blood streaks (affecting more than 5% but less than 30 % of the fibers seen at the surface of the dialyzer),
3b= More blood streaks (affecting more than 30% of the fibers seen at the surface if the dialyzer),
4=Complete occlusion


#### Appendix 16.2.5.9 Non-Study Producers (Safety Population)

| | | | | Proced | ure | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Dose Level/ | Subject | | Assessment | | | Due to Medical | Due to AE, | Overall Procedure | Procedure |
| Placebo | Number | Procedure | Date | Date | Time | History, seq# | AE page# | Interpretation | Findings/Comments |
| XXX <units></units> | X | None<br>XXXXXXXXXXXXX | DDMMYYYY | DDMMYYYY | HH:MM | XXXXXXX | XX | XXXXXXXXXXXXXXX | xxxxxxxxxxxxxx |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


#### Appendix 16.2.5.10 Prior and Concomitant Medications (Safety Population)

| | | | | | | | Start | | Stop | | | | | Prior | Due |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose Level/ | Subject | Any | Medication | Dosage/ | | | | | | | Fre- | | Con- | to | to |
| Placebo | Number | Med? | (WHO* Term) | Strength | Form | Route | Date | Time | Date | Time | quency | Indication | tinuing? | Study? | AE? |
| XXX <units></units> | X | No | None | | | | | | | | | | | | |
| | X | Yes | ACETAMINOPHEN | 620 mg/X | XXX | Oral | DDMMYYYY | HH:MM | DDMMYYYYY | HH:MM | Once | Toothache | No | X | XX |
| | | | (ACETAMINOPHEN) | _ | | | | | | | | | | | |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

Placebo = pooled placebo

\*Concomitant medications are coded with World Health Organization (WHO) Drug Dictionary Version September 2018, B3.

Med = Medication


#### Appendix 16.2.7.1.1 Adverse Events (I of II) (Safety Population)

| | | | | | Time From<br>Last Dose | Onset | | Resolve | d | Duration |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose Level/<br>Placebo | Subject<br>Number | TE?^ | Adverse Event* | Preferred Term | (DD:HH:MM) | Date | Time | Date | Time | (DD:HH:MM) |
| XXX <units></units> | X<br>X | Yes | None<br>XXXXXXXXXXXXX | *********** | xx:xx:xx | DDMMYYYY | XX:XX | DDMMYYYY | XX:XX | xx:xx:xx |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

Placebo = pooled placebo

\*Adverse events are classified according to MedDRA Version 21.1.

^TE = Treatment-emergent


#### Appendix 16.2.7.1.2 Adverse Events (II of II) (Safety Population)

| | | | | Onset | 5 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose Level/ | Subject | | Adverse | | | | Severity/ | | | Relationship to | |
| Placebo | Number | TE?^ | Event | Date | Time | Freq* | Intensity | Serious | Outcome | Study Drug | Action |
| XXX <units></units> | X | | None | | | | | | | | |
| | X | Yes | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMYYYY | XX:XX | Inter. | Grade 1<br>Mild | Not<br>serious | Resolved | XXXXXXXXXXXXXXX | XXXXXXXX |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3

Placebo = pooled placebo
^TE = Treatment-emergent

\*Freq represents Frequency: SI = Single Episode, Inter. = Intermittent, Cont. = Continuous


Appendix 16.2.7.2 Adverse Event Preferred Term Classification (Safety Population)

| | | | | | | Onset | |
|---|---|---|---|---|---|---|---|
| Dose Level/ | Subject | | Adverse | | | | |
| Placebo | Number | TE?^ | Event* | Preferred Term | System Organ Class | Date | Time |
| XXX <units></units> | X | Yes | XXXXXXX XXXXX XXXXX XXXXXX | XXXXXXXXX XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMYYYYY | XX:XX |

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo

\*Adverse events are classified according to MedDRA Version 21.1.

^TE = Treatment-emergent

#### Appendices 16.2.8.1.1 to 16.2.8.1.5 will have the following format.


Appendix 16.2.8.1.1 Clinical Laboratory Report - Serum Chemistry (Safety Population)

| Dose Level/ Subject<br>Placebo Number | Age#/<br>Sex | Study<br>Period Day | Hour | Date | Parameter1<br>< Range><br>(Unit) | Parameter2<br>< Range><br>(Unit) | Parameter3<br>< Range><br>(Unit) | Parameter4<br>< Range><br>(Unit) | Parameter5<br>< Range><br>(Unit) | Parameter6<br>< Range><br>(Unit) |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX <units> X</units> | XX/X | Screen .<br>X -X | -xx.x | DDMMMYYYY<br>DDMMMYYYY | XX H<br>XX L + | XX<br>XX L | XX<br>XX | XX<br>XX L | XX H<br>XX | XX<br>XX |

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early term chronologically with other scheduled assessments.

#### Programmer Note: All timepoints for coagulation and platelet count should be listed with results and flags.

```
Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3
0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3
Placebo = pooled placebo
#Age is calculated from the date of first dosing. F = Female; M = Male
H = Above reference range, L = Below reference range
PI interpretation: + = Clinically Significant
```


#### Appendix 16.2.8.2 Vital Signs (Safety Population)

| | | | | | | | Blood Pressure (mmHg) | | - | Tempera | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose Level/<br>Placebo | _ | Period | Day | Hour | Date | Time | Systolic/Diastolic | | ration<br>(bpm) | ture<br>(°C) | Weight<br>(kg) | Position |
| XXX <units></units> | X | Screen<br>XXX | - | -xx.x | DDMMYYYY<br>DDMMYYYYY | | <br>XXX/ XX<br>XXX/ XX | XX<br>XX | XX<br>XX | XX<br>XX | XX | XXXX |
| | | XXX | X | XX.X | DDMMYYYY | | XXX/ XX | XX | | | | |

Programmer Note: Sort unscheduled assessment and early term chronologically with other scheduled assessments.

Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3 0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3 Placebo = pooled placebo


Appendix 16.2.8.3 12-Lead Electrocardiogram (Safety Population)

| Dose Level/ Subject<br>Placebo Number | Period Day | Hour | Date | Time | Result | Heart<br>Rate<br>(bpm) | PR<br>(ms) | QRS<br>(ms) | QT<br>(ms) | QTcF*<br>(ms) | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX <units> X</units> | Screen .<br>X X<br>X X | XX.X<br>XX.X | | XX:XX | Normal<br>Normal | XX<br>XX<br>XX | XXX<br>XXX<br>XXX | XX<br>XX<br>XX | XXX<br>XXX<br>XXX | XXX^#<br>XXX<br>XXX | XXXXXXXXX |

Programmer Note: Sort unscheduled assessment and early term chronologically with other scheduled assessments.

```
Note: 0.25 mg/kg: Single IV Infusion of 0.25 mg/kg xisomab 3G3
0.5 mg/kg: Single IV Infusion of 0.5 mg/kg xisomab 3G3
Placebo = pooled placebo
QTcF* = QT corrected for heart rate using Fridericia's correction.
Abnormal, NCS = Abnormal, Not clinically significant
```

 $^{\circ}$  = QTcF is > 450 ms

# = QTcF change from baseline is > 30 ms